CLINICAL TRIAL: NCT02531802
Title: A Randomized, Double-blind, Placebo-controlled, Dose-Escalation Study Evaluating the Safety, Tolerability, and Immunogenicity of an Oral Inactivated ETEC Vaccine (ETVAX) Alone and Together With dmLT Adjuvant in Descending Age Groups in Bangladesh
Brief Title: Enterotoxigenic Escherichia Coli (ETEC) ETVAX Vaccine Trial in Bangladesh
Acronym: ETVAX/dmLT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: PATH (Other)
Collaborators: Scandinavian Biopharma AB (Industry); International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VAC 014
Record Dates: First submitted 2015-08-17; First posted 2015-08-24 (Estimated); Results first posted 2018-09-12 (Actual); Last update posted 2018-09-12 (Actual); Status verified 2018-09

CONDITIONS: Escherichia Coli Diarrhea
Keywords: ETEC diarrhea; Escherichia Coli (ETEC)
MeSH Terms: conditions — Escherichia coli Infections | interventions — Krebs-Ringer HEPES bicarbonate solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (21):
- Adult: ETVAX (Full) (Experimental): Adult arm (18-45 year olds) receiving the full dose of ETVAX vaccine (10^11 inactivated E. coli bacteria) added to bicarbonate buffer solution administered orally on Day 0 and 14
  Interventions: Biological: ETVAX; Other: Bicarbonate Buffer
- Adult: ETVAX (Full) + 10 ug dmLT (Experimental): Adult arm (18-45 year olds) receiving the full dose of ETVAX vaccine (10^11 inactivated E. coli bacteria) with 10 ug dmLT added to bicarbonate buffer solution administered orally on Day 0 and 14
  Interventions: Biological: ETVAX; Biological: dmLT; Other: Bicarbonate Buffer
- Adult: Placebo (Placebo Comparator): Adult arm (18-45 year olds) receiving a placebo on days 0 and 14
  Interventions: Other: Bicarbonate Buffer
- 24-59 months: ETVAX (1/4) (Experimental): 24-59 month old children receiving a quarter adult dose (2.5 x 10^10 inactivated E. coli bacteria) of ETVAX vaccine in bicarbonate buffer solution administered orally on Day 0 and 14
  Interventions: Biological: ETVAX; Other: Bicarbonate Buffer
- 24-59 months: ETVAX (1/2) (Experimental): 24-59 month old children receiving a half adult dose of ETVAX vaccine (5 x 10^10 inactivated E. coli bacteria) in bicarbonate buffer solution administered orally on Day 0 and 14
  Interventions: Biological: ETVAX; Other: Bicarbonate Buffer
- 24-59 months: ETVAX (full) (Experimental): 24-59 month old children receiving a full adult dose of ETVAX vaccine (10^11 inactivated E. coli bacteria) in bicarbonate buffer solution administered orally on Day 0 and 14
  Interventions: Biological: ETVAX; Other: Bicarbonate Buffer
- 24-59 months: ETVAX (1/2) + 2.5 ug dmLT (Experimental): 24-59 month old children receiving a half adult dose of ETVAX vaccine (5 x 10^10 inactivated E. coli bacteria) plus 2.5 ug dmLT in bicarbonate buffer solution administered orally on Day 0 and 14
  Interventions: Biological: ETVAX; Biological: dmLT; Other: Bicarbonate Buffer
- 24-59 months: ETVAX (1/2) + 5 ug dmLT (Experimental): 24-59 month old children receiving a half adult dose of ETVAX vaccine (5 x 10^10 inactivated E. coli bacteria) plus 5 ug dmLT in bicarbonate buffer solution administered orally on Day 0 and 14
  Interventions: Biological: ETVAX; Biological: dmLT; Other: Bicarbonate Buffer
- 24-59 months: ETVAX (1/2) + 10 ug dmLT (Experimental): 24-59 month old children receiving a half adult dose of ETVAX vaccine (5 x 10^10 inactivated E. coli bacteria) plus 10 ug dmLT in bicarbonate buffer solution administered orally on Day 0 and 14
  Interventions: Biological: ETVAX; Biological: dmLT; Other: Bicarbonate Buffer
- 24-59 months: Placebo (Placebo Comparator): 24-59 month old children receiving a placebo of bicarbonate buffer solution administered orally on Day 0 and 14
  Interventions: Other: Bicarbonate Buffer
- 12-23 months: ETVAX (1/4) (Experimental): 12-23 month old children receiving a quarter adult dose of ETVAX vaccine (2.5 x 10^10 inactivated E. coli bacteria) in bicarbonate buffer solution administered orally on Day 0 and 14
  Interventions: Biological: ETVAX; Other: Bicarbonate Buffer
- 12-23 months: ETVAX (1/2) (Experimental): 12-23 month old children receiving a half adult dose of ETVAX vaccine (5 x 10^10 inactivated E. coli bacteria) in bicarbonate buffer solution administered orally on Day 0 and 14
  Interventions: Biological: ETVAX; Other: Bicarbonate Buffer
- 12-23 months: ETVAX (1/2) + 2.5 ug dmLT (Experimental): 12-23 month old children receiving a half adult dose of ETVAX vaccine (5 x 10^10 inactivated E. coli bacteria) plus 2.5 ug dmLT in bicarbonate buffer solution administered orally on Day 0 and 14
  Interventions: Biological: ETVAX; Biological: dmLT; Other: Bicarbonate Buffer
- 12-23 months: ETVAX (1/2) + 5 ug dmLT (Experimental): 12-23 month old children receiving a half adult dose of ETVAX vaccine (5 x 10^10 inactivated E. coli bacteria) plus 5 ug dmLT in bicarbonate buffer solution administered orally on Day 0 and 14
  Interventions: Biological: ETVAX; Biological: dmLT; Other: Bicarbonate Buffer
- 12-23 months: Placebo (Placebo Comparator): 12-23 month old children receiving a placebo of bicarbonate buffer solution administered orally on Day 0 and 14
  Interventions: Other: Bicarbonate Buffer
- 6-11 months: ETVAX (1/8) (Experimental): 6-11 month old children receiving an eighth of an adult dose of ETVAX vaccine in bicarbonate buffer solution administered orally on Day 0 and 14
  Interventions: Biological: ETVAX; Other: Bicarbonate Buffer
- 6-11 months: ETVAX (1/4) (Experimental): 6-11 month old children receiving a quarter of an adult dose of ETVAX vaccine (2.5 x 10^10 inactivated E. coli bacteria) in bicarbonate buffer solution administered orally on Day 0 and 14
  Interventions: Biological: ETVAX; Other: Bicarbonate Buffer
- 6-11 months: ETVAX (1/2) (Experimental): 6-11 month old children receiving a half of an adult dose of ETVAX vaccine (5 x 10^10 inactivated E. coli bacteria) in bicarbonate buffer solution administered orally on Day 0 and 14
  Interventions: Biological: ETVAX; Other: Bicarbonate Buffer
- 6-11 months: ETVAX (1/4) + 2.5 ug dmLT (Experimental): 6-11 month old children receiving a quarter of an adult dose of ETVAX vaccine (2.5 x 10^10 inactivated E. coli bacteria) plus 2.5 ug dmLT in bicarbonate buffer solution administered orally on Day 0 and 14
  Interventions: Biological: ETVAX; Biological: dmLT; Other: Bicarbonate Buffer
- 6-11 month olds: ETVAX (1/4) + 5 ug dmLT (Experimental): 6-11 month old children receiving a quarter of an adult dose of ETVAX vaccine (2.5 x 10^10 inactivated E. coli bacteria) plus 5 ug dmLT in bicarbonate buffer solution administered orally on Day 0 and 14
  Interventions: Biological: ETVAX; Biological: dmLT; Other: Bicarbonate Buffer
- 6-11 month olds: Placebo (Placebo Comparator): 6-11 month old children receiving a placebo of bicarbonate buffer solution administered orally on Day 0 and 14
  Interventions: Other: Bicarbonate Buffer

INTERVENTIONS:
Biological: ETVAX — Varying dosages of liquid ETVAX vaccine (Batch BX1003574). A full dose consisted of:
  * Hybrid protein between the B-subunit of the E. coli heat-labile enterotoxin and the B-subunit of the cholera toxin (LCTBA): 1 mg
  * E. coli ETEX 21 formalin inactivated: 1.3 mg colonization factor 1 (CFA/I)
  * E. coli ETEX 22 formalin inactivated: 6.4 mg coli surface antigen 3 (CS3)
  * E. coli ETEX 23 formalin inactivated: 1.1 mg coli surface antigen 5 (CS5)
  * E. coli ETEX 24 phenol inactivated: 0.5 mg coli surface antigen 6 (CS6)
  The vaccine was given together with sodium bicarbonate effervescent granules (Recip), which was dissolved in water and mixed with the vaccine suspension prior to oral administration. The buffer was used to prevent degradation of LCTBA hybrid protein by the gastric acid.
  Arms: 12-23 months: ETVAX (1/2); 12-23 months: ETVAX (1/2) + 2.5 ug dmLT; 12-23 months: ETVAX (1/2) + 5 ug dmLT; 12-23 months: ETVAX (1/4); 24-59 months: ETVAX (1/2); 24-59 months: ETVAX (1/2) + 10 ug dmLT; 24-59 months: ETVAX (1/2) + 2.5 ug dmLT; 24-59 months: ETVAX (1/2) + 5 ug dmLT; 24-59 months: ETVAX (1/4); 24-59 months: ETVAX (full); 6-11 month olds: ETVAX (1/4) + 5 ug dmLT; 6-11 months: ETVAX (1/2); 6-11 months: ETVAX (1/4); 6-11 months: ETVAX (1/4) + 2.5 ug dmLT; 6-11 months: ETVAX (1/8); Adult: ETVAX (Full); Adult: ETVAX (Full) + 10 ug dmLT
Biological: dmLT — Varying dosages of dmLT, a derivative of wild-type enterotoxigenic Escherichia coli LT that has been genetically modified by replacing the arginine at amino acid position 192 with glycine and the leucine at amino acid position 211 with alanine. These two amino acid substitutions take place in proteolytic cleavage sites which are critical for activation of the secreted toxin molecules.
  Other Names: double mutant heat labile toxin, LT(R192G/L211A)
  Arms: 12-23 months: ETVAX (1/2) + 2.5 ug dmLT; 12-23 months: ETVAX (1/2) + 5 ug dmLT; 24-59 months: ETVAX (1/2) + 10 ug dmLT; 24-59 months: ETVAX (1/2) + 2.5 ug dmLT; 24-59 months: ETVAX (1/2) + 5 ug dmLT; 6-11 month olds: ETVAX (1/4) + 5 ug dmLT; 6-11 months: ETVAX (1/4) + 2.5 ug dmLT; Adult: ETVAX (Full) + 10 ug dmLT
Other: Bicarbonate Buffer — Sodium bicarbonate buffer dissolved in 150 ml of potable water

SUMMARY:
The purpose of this study is to determine if the ETEC vaccine ETVAX with and without dmLT adjuvant is safe and immunogenic in adults, children, toddlers and infants in Bangladesh.

DETAILED DESCRIPTION:
This Phase I/II trial will serve to assess whether ETVAX is safe and provides mucosal as well as systemic immune responses against the key protective antigens when tested in different age-groups in Bangladesh. This study provides an opportunity to test the safety profile of a mucosal adjuvant, double-mutant LT (dmLT), in adults and children, as well as provide the opportunity to potentially assess the ability of dmLT to further enhance the mucosal and systemic antibody responses to key antigens in the ETVAX vaccine among age groups in developing country sites, like Bangladesh, that have proved refractory to oral immunization with enteric vaccines. In addition, this study also allows for the evaluation of the potential dose-sparing effect of dmLT when combined with a lower dose of vaccine. Finally, this clinical trial is considered an essential study along the critical path of the overall clinical development plan before determining whether the vaccine can be tested for protective efficacy in children in developing countries.

ELIGIBILITY:
Adults

Inclusion Criteria:

1. Healthy male or female adults 18-45 years old, inclusive
2. General good health as determined by the screening evaluation no greater than 7days before enrollment and vaccination
3. Properly informed about the study, able to understand it and sign or thumb print the informed consent form
4. Available for the entire period of the study and reachable by study staff throughout the entire follow-up period
5. Females of childbearing potential who are willing to take a urine pregnancy test at screening and before the second vaccination. Pregnancy tests must be negative before each vaccination. Females of childbearing potential must agree to use an efficacious hormonal or barrier method of birth control during the study. Abstinence is also acceptable.
6. Informed Consent (signature or thumb print provided, with witness signature)

Exclusion Criteria:

1. Presence of any significant known systemic disorder (cardiovascular, pulmonary, hepatic, renal, gastrointestinal, endocrine, immunological, dermatological, neurological, cancer or autoimmune disease) as determined by medical history and/or physical examination which would endanger the participant's health or is likely to result in non-conformance to the protocol.
2. History of congenital abdominal disorders, intussusception, abdominal surgery or any other congenital disorder or presence of a significant medical condition that in the opinion of the Investigator precludes participation in the study. Known or suspected impairment of immunological function based on medical history and physical examination. Clinical evidence of active gastrointestinal illness and acute disease at the time of enrollment
3. Screening positive with hepatitis B antigen and/or hepatitis C antibodies
4. Participation in research involving another investigational product (defined as receipt of investigational product) during the 30 days before planned date of first vaccination or concurrently participating in another clinical study at any time during the study period, in which the participant has been or will be exposed to an investigational or a non-investigational product
5. Clinically significant abnormalities in screening hematology or serum chemistry, as determined by the Study Physician
6. History of febrile illness within 48 hours prior to vaccination and fever at the time of immunization (fever is defined as a temperature ≥ 37.5 C (99.5 F) on axillary, oral, or tympanic measurement)
7. Prior receipt of any cholera (e.g., Dukoral, Shanchol) or ETEC vaccine
8. Prior receipt of a blood transfusion or blood products, including immunoglobulins
9. Evidence of current illicit drug use or drug dependence
10. Current use of iron or zinc supplements within the past 7 days; current use of antacids (H2 blockers, omeprazole, over-the-counter (OTC) agents) or immunosuppressive drug
11. Any condition which, in the opinion of the investigator, might jeopardize the safety of study participants or interfere with the evaluation of the study objectives
12. Receipt of antimicrobial drugs for any reason within 14 days before vaccination
13. History of diarrhea during the 7 days before vaccination (see protocol definition of diarrhea)
14. Culture positive for ETEC, Shigella, V. Cholerae or Salmonella within 7 days before vaccination.
15. Acute disease at the time of enrollment or 3 days prior to enrollment
16. History of chronic administration (defined as more than 14 days) of immunosuppressant medications, including corticosteroids.

Children, Toddlers and Infants Inclusion Criteria

1. Healthy male or female infants/toddlers/children ages:

   * Part B: >24 and ≤59 months old at the time of enrollment
   * Part C: ≥12 and <24 months old at the time of enrollment
   * Part D: ≥6 and <12 months at the time of enrollment
2. General good health as determined by the screening evaluation no greater than 7 days before enrollment and vaccination
3. Parent properly informed about the study, able to understand it and sign or thumb print the informed consent form
4. Parent and child available for the entire study period of the study and reachable by study staff throughout the entire follow-up period
5. Informed Consent (signature or thumb of parent, with signature of witness, provided)

Exclusion Criteria

1. Presence of any significant known systemic disorder (cardiovascular, pulmonary, hepatic, renal, gastrointestinal, endocrine, immunological, dermatological, neurological, cancer or autoimmune disease) as determined by medical history and/or physical examination which would endanger the participant's health or is likely to result in non-conformance to the protocol.
2. History of congenital abdominal disorders, intussusception, abdominal surgery or any other congenital disorder or presence of a significant medical condition that in the opinion of the Investigator precludes participation in the study. Known or suspected impairment of immunological function based on medical history and physical examination. Clinical evidence of active gastrointestinal illness and acute disease at the time of enrollment
3. Screening positive with hepatitis B antigen and/or hepatitis C antibodies
4. Participation in research involving another investigational product (defined as receipt of investigational product) during the 30 days before planned date of first vaccination or concurrently participating in another clinical study at any time during the study period, in which the participant has been or will be exposed to an investigational or a non-investigational product
5. Clinically significant abnormalities in screening hematology or serum chemistry, as determined by the Study Physician
6. History of febrile illness within 48 hours prior to vaccination and fever at the time of immunization (fever is defined as a temperature ≥ 37.5 C (99.5 F) on axillary, oral, or tympanic measurement)
7. Prior receipt of any cholera (e.g., Dukoral, Shanchol) or ETEC vaccine
8. Prior receipt of a blood transfusion or blood products, including immunoglobulins
9. Current use of iron or zinc supplements within the past 7 days; current use of antacids (H2 blockers, omeprazole, OTC agents) or immunosuppressive drug
10. Any condition which, in the opinion of the investigator, might jeopardize the safety of study participants or interfere with the evaluation of the study objectives
11. Receipt of antimicrobial drugs for any reason within 14 days before vaccination
12. History of diarrhea during the 7 days before vaccination (see Protocol definition of diarrhea))
13. Culture positive for ETEC, Shigella, V. cholerae, Salmonella or Rotavirus (the latter for all children <5 years of age) within 7 days of vaccination
14. Acute disease at the time of enrollment or 3 days prior to enrollment
15. Known or suspected impairment of immunological function based on medical history and physical examination
16. Participant's parents/guardians not able, available or willing to accept active weekly follow-up by the study staff
17. History of chronic administration (defined as more than 14 days) of immunosuppressant medications, including corticosteroids. Infants on inhaled or topical steroids may be permitted to participate in the study
18. Any medical condition in the child/infant that, in the judgment of the investigator, would interfere with or serves as a contraindication to protocol adherence or a participant's parents' ability to give informed consent
19. Medically significant malnutrition, defined as moderate malnutrition (wt-for-ht z-score between -3.0 and -2.0) and severe malnutrition (wt-for-ht z-score <-3.0 or edema)

Ages: 6 Months to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 475 (Actual)
Dates: Start 2015-10; Primary Completion 2017-07-29 (Actual); Study Completion 2017-07-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- International Centre for Diarrheal Disease, Bangladesh (icddr,b), Dhaka, Bangladesh

REFERENCES:
- [Derived] Higginson EE, Sayeed MA, Pereira Dias J, Shetty V, Ballal M, Srivastava SK, Willis I, Qadri F, Dougan G, Mutreja A. Microbiome Profiling of Enterotoxigenic Escherichia coli (ETEC) Carriers Highlights Signature Differences between Symptomatic and Asymptomatic Individuals. mBio. 2022 Jun 28;13(3):e0015722. doi: 10.1128/mbio.00157-22. Epub 2022 May 10. PMID 35536001
- [Derived] Qadri F, Akhtar M, Bhuiyan TR, Chowdhury MI, Ahmed T, Rafique TA, Khan A, Rahman SIA, Khanam F, Lundgren A, Wiklund G, Kaim J, Lofstrand M, Carlin N, Bourgeois AL, Maier N, Fix A, Wierzba T, Walker RI, Svennerholm AM. Safety and immunogenicity of the oral, inactivated, enterotoxigenic Escherichia coli vaccine ETVAX in Bangladeshi children and infants: a double-blind, randomised, placebo-controlled phase 1/2 trial. Lancet Infect Dis. 2020 Feb;20(2):208-219. doi: 10.1016/S1473-3099(19)30571-7. Epub 2019 Nov 19. PMID 31757774
- [Derived] Akhtar M, Chowdhury MI, Bhuiyan TR, Kaim J, Ahmed T, Rafique TA, Khan A, Rahman SIA, Khanam F, Begum YA, Sharif MZ, Islam LN, Carlin N, Maier N, Fix A, Wierzba TF, Walker RI, Bourgeois AL, Svennerholm AM, Qadri F, Lundgren A. Evaluation of the safety and immunogenicity of the oral inactivated multivalent enterotoxigenic Escherichia coli vaccine ETVAX in Bangladeshi adults in a double-blind, randomized, placebo-controlled Phase I trial using electrochemiluminescence and ELISA assays for immunogenicity analyses. Vaccine. 2019 Sep 3;37(37):5645-5656. doi: 10.1016/j.vaccine.2018.11.040. Epub 2018 Nov 22. PMID 30473185

RESULTS

PARTICIPANT FLOW:
Period: Received Vaccination 1
Arm/Group | Adult: ETVAX (Full) | Adult: ETVAX (Full) + 10 ug dmLT | Adult: Placebo | 24-59 Months: ETVAX (1/4) | 24-59 Months: ETVAX (1/2) | 24-59 Months: ETVAX (Full) | 24-59 Months: ETVAX (1/2) + 2.5 ug dmLT | 24-59 Months: ETVAX (1/2) + 5 ug dmLT | 24-59 Months: ETVAX (1/2) + 10 ug dmLT | 24-59 Months: Placebo | 12-23 Months: ETVAX (1/4) | 12-23 Months: ETVAX (1/2) | 12-23 Months: ETVAX (1/2) + 2.5 ug dmLT | 12-23 Months: ETVAX (1/2) + 5 ug dmLT | 12-23 Months: Placebo | 6-11 Months: ETVAX (1/8) | 6-11 Months: ETVAX (1/4) | 6-11 Months: ETVAX (1/2) | 6-11 Months: ETVAX (1/4) + 2.5 ug dmLT | 6-11 Month Olds: ETVAX (1/4) + 5 ug dmLT | 6-11 Month Olds: Placebo
Started | 15 | 15 | 15 | 15 | 15 | 3 | 15 | 15 | 15 | 52 | 15 | 15 | 15 | 15 | 40 | 30 | 30 | 30 | 30 | 30 | 50
Completed | 15 | 15 | 15 | 15 | 15 | 3 | 15 | 15 | 15 | 52 | 15 | 15 | 15 | 15 | 40 | 30 | 30 | 30 | 30 | 30 | 50
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Received Vaccination 2
Arm/Group | Adult: ETVAX (Full) | Adult: ETVAX (Full) + 10 ug dmLT | Adult: Placebo | 24-59 Months: ETVAX (1/4) | 24-59 Months: ETVAX (1/2) | 24-59 Months: ETVAX (Full) | 24-59 Months: ETVAX (1/2) + 2.5 ug dmLT | 24-59 Months: ETVAX (1/2) + 5 ug dmLT | 24-59 Months: ETVAX (1/2) + 10 ug dmLT | 24-59 Months: Placebo | 12-23 Months: ETVAX (1/4) | 12-23 Months: ETVAX (1/2) | 12-23 Months: ETVAX (1/2) + 2.5 ug dmLT | 12-23 Months: ETVAX (1/2) + 5 ug dmLT | 12-23 Months: Placebo | 6-11 Months: ETVAX (1/8) | 6-11 Months: ETVAX (1/4) | 6-11 Months: ETVAX (1/2) | 6-11 Months: ETVAX (1/4) + 2.5 ug dmLT | 6-11 Month Olds: ETVAX (1/4) + 5 ug dmLT | 6-11 Month Olds: Placebo
Started | 15 | 15 | 15 | 15 | 15 | 3 | 15 | 15 | 15 | 52 | 15 | 15 | 15 | 15 | 40 | 30 | 30 | 30 | 30 | 30 | 50
Completed | 15 | 15 | 14 | 15 | 15 | 0 | 15 | 15 | 15 | 49 | 13 | 15 | 13 | 13 | 39 | 30 | 30 | 26 | 27 | 29 | 49
Not Completed | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 3 | 2 | 0 | 2 | 2 | 1 | 0 | 0 | 4 | 3 | 1 | 1
Not completed — Medication interfering with study taken | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adult: Placebo | Adult: ETVAX (Full) | Adult: ETVAX (Full) + 10 ug dmLT | 24-59 Months: Placebo | 24-59 Months: ETVAX (1/4) | 24-59 Months: ETVAX (1/2) | 24-59 Months: ETVAX (Full) | 24-59 Months: ETVAX (1/2) + 2.5 ug dmLT | 24-59 Months: ETVAX (1/2) + 5 ug dmLT | 24-59 Months: ETVAX (1/2) + 10 ug dmLT | 12-23 Months: Placebo | 12-23 Months: ETVAX (1/4) | 12-23 Months: ETVAX (1/2) | 12-23 Months: ETVAX (1/2) + 2.5 ug dmLT | 12-23 Months: ETVAX (1/2) + 5 ug dmLT | 6-11 Month Olds: Placebo | 6-11 Months: ETVAX (1/8) | 6-11 Months: ETVAX (1/4) | 6-11 Months: ETVAX (1/2) | 6-11 Months: ETVAX (1/4) + 2.5 ug dmLT | 6-11 Month Olds: ETVAX (1/4) + 5 ug dmLT | Total
Number analyzed (Participants) | 15 | 15 | 15 | 52 | 15 | 15 | 3 | 15 | 15 | 15 | 40 | 15 | 15 | 15 | 15 | 50 | 30 | 30 | 30 | 30 | 30 | 475
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.5 (5.58) | 30.1 (6.96) | 29.4 (6.96) | 3.7 (0.77) | 4.1 (0.62) | 3.4 (0.68) | 4.2 (0.59) | 3.4 (0.86) | 3.6 (0.91) | 3.4 (0.73) | 1.4 (0.27) | 1.3 (0.21) | 1.5 (0.30) | 1.6 (0.28) | 1.4 (0.27) | 0.7 (0.13) | 0.7 (0.15) | 0.7 (0.14) | 0.7 (0.11) | 0.7 (0.15) | 0.6 (0.10) | 4.4 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 11 | 26 | 10 | 6 | 2 | 6 | 7 | 9 | 20 | 6 | 5 | 7 | 10 | 23 | 14 | 19 | 16 | 18 | 16 | 249
  Male | 5 | 7 | 4 | 26 | 5 | 9 | 1 | 9 | 8 | 6 | 20 | 9 | 10 | 8 | 5 | 27 | 16 | 11 | 14 | 12 | 14 | 226
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 15 | 15 | 15 | 52 | 15 | 15 | 3 | 15 | 15 | 15 | 40 | 15 | 15 | 15 | 15 | 50 | 30 | 30 | 30 | 30 | 30 | 475
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Height [Mean (Standard Deviation); unit: centimeters] | 154.69 (8.01) | 155.29 (9.38) | 154.26 (10.16) | 97.02 (6.84) | 97.73 (5.33) | 93.73 (7.08) | 96.67 (2.52) | 90.33 (6.11) | 94.13 (7.27) | 92.2 (6.59) | 77.83 (4.60) | 76.27 (2.99) | 79.33 (4.27) | 79.2 (4.69) | 76.6 (2.59) | 67.64 (3.44) | 68.83 (3.04) | 67.77 (3.45) | 68.83 (3.04) | 66.73 (3.14) | 67.57 (2.58) | 85.6 (25.6)
Weight [Mean (Standard Deviation); unit: kilograms] | 56.65 (9.867) | 56.86 (11.776) | 55.25 (11.441) | 13.71 (2.043) | 13.59 (1.488) | 13.61 (1.914) | 12.43 (0.513) | 12.1 (1.465) | 13.35 (1.957) | 12.61 (1.936) | 9.47 (1.226) | 9.23 (0.959) | 9.64 (0.946) | 9.5 (1.271) | 9.24 (0.998) | 7.66 (0.958) | 7.84 (1.006) | 7.37 (0.728) | 7.85 (1.226) | 7.41 (0.876) | 7.76 (0.598) | 14.2 (14.3)

OUTCOME MEASURES:

1. Primary Outcome: Number and Percentage of Participants Experiencing Solicited Events by Symptom and Maximum Severity
Description: Adverse events (AEs) were assessed post-vaccination using participant/parent/guardian interview (including memory aids), targeted physical examinations, vital signs and clinical laboratory tests and reactogenicity assessments which were completed following each vaccination. The solicited AEs of nausea (adults only), abdominal pain/stomach ache (adults and children 24-59 months only), fever, vomiting and diarrhea were evaluated daily for 7 days post vaccination.
Time Frame: 7 days after each vaccination (Day 7 and Day 21)
Measure: Count of Participants; unit: Participants
Arm/Group | Adult: ETVAX (Full) | Adult: ETVAX (Full) + 10 ug dmLT | Adult: Placebo | 24-59 Months: ETVAX (1/4) | 24-59 Months: ETVAX (1/2) | 24-59 Months: ETVAX (Full) | 24-59 Months: ETVAX (1/2) + 2.5 ug dmLT | 24-59 Months: ETVAX (1/2) + 5 ug dmLT | 24-59 Months: ETVAX (1/2) + 10 ug dmLT | 24-59 Months: Placebo | 12-23 Months: ETVAX (1/4) | 12-23 Months: ETVAX (1/2) | 12-23 Months: ETVAX (1/2) + 2.5 ug dmLT | 12-23 Months: ETVAX (1/2) + 5 ug dmLT | 12-23 Months: Placebo | 6-11 Months: ETVAX (1/8) | 6-11 Months: ETVAX (1/4) | 6-11 Months: ETVAX (1/2) | 6-11 Months: ETVAX (1/4) + 2.5 ug dmLT | 6-11 Month Olds: ETVAX (1/4) + 5 ug dmLT | 6-11 Month Olds: Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15 | 3 | 15 | 15 | 15 | 52 | 15 | 15 | 15 | 15 | 40 | 30 | 30 | 30 | 30 | 30 | 50
Participants
  Elevated oral temperature: None | 15 | 14 | 15 | 15 | 14 | 3 | 12 | 15 | 15 | 50 | 14 | 15 | 12 | 14 | 39 | 28 | 28 | 28 | 28 | 27 | 48
  Elevated oral temperature: Mild | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 2 | 1 | 1 | 2 | 2 | 1 | 2 | 3 | 2
  Elevated oral temperature: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Vomiting: None | 15 | 15 | 15 | 13 | 15 | 1 | 13 | 14 | 12 | 52 | 13 | 14 | 13 | 7 | 40 | 28 | 25 | 20 | 23 | 25 | 48
  Vomiting: Mild | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 3 | 0 | 2 | 1 | 2 | 8 | 0 | 2 | 5 | 8 | 6 | 5 | 2
  Vomiting: Moderate | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
  Loose stools: None | 15 | 15 | 15 | 15 | 15 | 3 | 15 | 15 | 15 | 52 | 15 | 15 | 12 | 15 | 40 | 30 | 29 | 29 | 30 | 30 | 50
  Loose stools: Mild | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
  Loose stools: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Abdominal pain/stomach ache: None | 15 | 15 | 15 | 15 | 15 | 3 | 15 | 15 | 15 | 52 | 15 | 15 | 15 | 15 | 40 | 30 | 30 | 30 | 30 | 30 | 50
  Abdominal pain/stomach ache: Mild | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Abdominal pain/stomach ache: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Diarrhea: None | 15 | 15 | 15 | 15 | 15 | 3 | 15 | 15 | 15 | 52 | 14 | 14 | 15 | 14 | 40 | 30 | 30 | 28 | 29 | 29 | 50
  Diarrhea: Mild | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 1 | 0
  Diarrhea: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Acute systemic allergic reaction: None | 15 | 15 | 15 | 15 | 15 | 3 | 15 | 15 | 15 | 52 | 15 | 15 | 15 | 15 | 40 | 30 | 30 | 30 | 30 | 30 | 50
  Acute systemic allergic reaction: Mild | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Acute systemic allergic reaction: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Nausea: None | 15 | 15 | 15 | 15 | 15 | 3 | 15 | 15 | 15 | 52 | 15 | 15 | 15 | 15 | 40 | 30 | 30 | 30 | 30 | 30 | 50
  Nausea: Mild | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Nausea: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any symptom: None | 15 | 14 | 15 | 13 | 14 | 1 | 11 | 14 | 12 | 50 | 12 | 13 | 9 | 7 | 40 | 26 | 23 | 17 | 22 | 22 | 46
  Any symptom: Mild | 0 | 1 | 0 | 2 | 1 | 0 | 3 | 0 | 3 | 2 | 2 | 2 | 5 | 8 | 0 | 4 | 7 | 10 | 7 | 8 | 4
  Any symptom: Moderate | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0

2. Primary Outcome: Number and Percentage of Participants Experiencing Unsolicited Adverse Events Related to Vaccine
Description: Adverse events (AEs) were assessed post-vaccination using participant/parent/guardian interview (including memory aids), targeted physical examinations, vital signs and clinical laboratory tests and reactogenicity assessments which were completed following each vaccination. Unsolicited AEs were assessed through Day 42 and serious adverse events (SAEs) were assessed over the entire duration of the study.
Time Frame: 6 months ± 14 days after the first dose
Measure: Count of Participants; unit: Participants
Arm/Group | Adult: ETVAX (Full) | Adult: ETVAX (Full) + 10 ug dmLT | Adult: Placebo | 24-59 Months: ETVAX (1/4) | 24-59 Months: ETVAX (1/2) | 24-59 Months: ETVAX (Full) | 24-59 Months: ETVAX (1/2) + 2.5 ug dmLT | 24-59 Months: ETVAX (1/2) + 5 ug dmLT | 24-59 Months: ETVAX (1/2) + 10 ug dmLT | 24-59 Months: Placebo | 12-23 Months: ETVAX (1/4) | 12-23 Months: ETVAX (1/2) | 12-23 Months: ETVAX (1/2) + 2.5 ug dmLT | 12-23 Months: ETVAX (1/2) + 5 ug dmLT | 12-23 Months: Placebo | 6-11 Months: ETVAX (1/8) | 6-11 Months: ETVAX (1/4) | 6-11 Months: ETVAX (1/2) | 6-11 Months: ETVAX (1/4) + 2.5 ug dmLT | 6-11 Month Olds: ETVAX (1/4) + 5 ug dmLT | 6-11 Month Olds: Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15 | 3 | 15 | 15 | 15 | 52 | 15 | 15 | 15 | 15 | 40 | 30 | 30 | 30 | 30 | 30 | 50
Participants
  Leukocytosis: Mild | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytosis: Moderate | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytosis: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytosis: No AE related to vaccine | 15 | 14 | 15 | 15 | 15 | 3 | 15 | 15 | 15 | 52 | 14 | 15 | 14 | 15 | 38 | 30 | 30 | 30 | 30 | 30 | 50
  Alanine aminotransferase increased: Mild | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Alanine aminotransferase increased: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Alanine aminotransferase increased: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Alanine aminotransferase increased: No AE related to vaccine | 15 | 15 | 15 | 15 | 15 | 3 | 15 | 15 | 15 | 52 | 15 | 15 | 15 | 15 | 39 | 30 | 30 | 30 | 30 | 30 | 49

3. Secondary Outcome: Number and Percentage of Subjects With ≥Two-fold Increase in Antibody Lymphocyte Supernatant (ALS) Immunoglobulin A (IgA) Response After Either Vaccine Dose, by Antigen
Description: Between baseline and post-immunization (measured 7 days after the first dose and 5 days after the second). Antigen in ETVAX were:
  E. coli, CFA/I, strain ETEX 21 formalin inactivated, E. coli, CS3, strain ETEX 22 formalin inactivated, E. coli, CS5, strain ETEX 23 formalin inactivated, E. coli, CS6, strain ETEX 24 phenol inactivated, B-subunit of the E. coli heat-labile enterotoxin
Time Frame: 19 days
Population: Subjects who received both vaccinations and had valid baseline and endline immunologic samples.
Measure: Count of Participants; unit: Participants
Arm/Group | Adult: ETVAX (Full) | Adult: ETVAX (Full) + 10 ug dmLT | Adult: Placebo | 24-59 Months: ETVAX (1/4) | 24-59 Months: ETVAX (1/2) | 24-59 Months: ETVAX (1/2) + 2.5 ug dmLT | 24-59 Months: ETVAX (1/2) + 5 ug dmLT | 24-59 Months: ETVAX (1/2) + 10 ug dmLT | 24-59 Months: Placebo | 12-23 Months: ETVAX (1/4) | 12-23 Months: ETVAX (1/2) | 12-23 Months: ETVAX (1/2) + 2.5 ug dmLT | 12-23 Months: ETVAX (1/2) + 5 ug dmLT | 12-23 Months: Placebo | 6-11 Months: ETVAX (1/8) | 6-11 Months: ETVAX (1/4) | 6-11 Months: ETVAX (1/2) | 6-11 Months: ETVAX (1/4) + 2.5 ug dmLT | 6-11 Month Olds: ETVAX (1/4) + 5 ug dmLT | 6-11 Month Olds: Placebo
Number analyzed (Participants) | 15 | 15 | 14 | 15 | 15 | 15 | 15 | 15 | 49 | 13 | 15 | 13 | 13 | 39 | 30 | 30 | 24 | 26 | 29 | 49
Participants
  CFA/I: Yes | 15 | 15 | 0 | 15 | 14 | 15 | 14 | 13 | 3 | 11 | 11 | 9 | 9 | 3 | 15 | 9 | 12 | 10 | 7 | 7
  CFA/I: No | 0 | 0 | 14 | 0 | 1 | 0 | 1 | 2 | 46 | 2 | 4 | 4 | 4 | 36 | 15 | 21 | 12 | 16 | 22 | 42
  CS3: Yes | 15 | 15 | 4 | 15 | 14 | 15 | 13 | 15 | 7 | 11 | 13 | 12 | 7 | 6 | 15 | 13 | 13 | 13 | 11 | 8
  CS3: No | 0 | 0 | 10 | 0 | 1 | 0 | 2 | 0 | 42 | 2 | 2 | 1 | 6 | 33 | 15 | 17 | 11 | 13 | 18 | 41
  CS5: Yes | 15 | 15 | 0 | 14 | 13 | 12 | 12 | 11 | 2 | 8 | 7 | 6 | 8 | 3 | 11 | 6 | 5 | 5 | 3 | 7
  CS5: No | 0 | 0 | 14 | 1 | 2 | 3 | 3 | 4 | 47 | 5 | 8 | 7 | 5 | 36 | 19 | 24 | 19 | 21 | 26 | 42
  CS6: number analyzed (Participants) | 15 | 15 | 14 | 15 | 15 | 15 | 15 | 15 | 49 | 12 | 15 | 13 | 13 | 39 | 30 | 30 | 24 | 26 | 29 | 49
  CS6: Yes | 15 | 15 | 1 | 12 | 12 | 14 | 12 | 10 | 1 | 6 | 5 | 9 | 5 | 5 | 3 | 5 | 5 | 0 | 0 | 2
  CS6: No | 0 | 0 | 13 | 3 | 3 | 1 | 3 | 5 | 48 | 6 | 10 | 4 | 8 | 34 | 27 | 25 | 19 | 26 | 29 | 47
  LTB: Yes | 15 | 15 | 0 | 15 | 15 | 15 | 15 | 15 | 4 | 13 | 15 | 13 | 11 | 6 | 19 | 24 | 20 | 18 | 21 | 15
  LTB: No | 0 | 0 | 14 | 0 | 0 | 0 | 0 | 0 | 45 | 0 | 0 | 0 | 2 | 33 | 11 | 6 | 4 | 8 | 8 | 34

4. Secondary Outcome: Number and Percentage of Subjects With ≥Four-fold Increase in Antibody Lymphocyte Supernatant (ALS) Immunoglobulin A (IgA) Response After Either Vaccine Dose, by Antigen
Description: as for outcome 3
Time Frame: 19 days
Population: Subjects who received both vaccinations and had valid baseline and endline immunologic samples.
Measure: Count of Participants; unit: Participants
Arm/Group | Adult: ETVAX (Full) | Adult: ETVAX (Full) + 10 ug dmLT | Adult: Placebo | 24-59 Months: ETVAX (1/4) | 24-59 Months: ETVAX (1/2) | 24-59 Months: ETVAX (1/2) + 2.5 ug dmLT | 24-59 Months: ETVAX (1/2) + 5 ug dmLT | 24-59 Months: ETVAX (1/2) + 10 ug dmLT | 24-59 Months: Placebo | 12-23 Months: ETVAX (1/4) | 12-23 Months: ETVAX (1/2) | 12-23 Months: ETVAX (1/2) + 2.5 ug dmLT | 12-23 Months: ETVAX (1/2) + 5 ug dmLT | 12-23 Months: Placebo | 6-11 Months: ETVAX (1/8) | 6-11 Months: ETVAX (1/4) | 6-11 Months: ETVAX (1/2) | 6-11 Months: ETVAX (1/4) + 2.5 ug dmLT | 6-11 Month Olds: ETVAX (1/4) + 5 ug dmLT | 6-11 Month Olds: Placebo
Number analyzed (Participants) | 15 | 15 | 14 | 15 | 15 | 15 | 15 | 15 | 49 | 13 | 15 | 13 | 13 | 39 | 30 | 30 | 24 | 26 | 29 | 49
Participants
  CFA/I: Yes | 15 | 15 | 0 | 15 | 12 | 14 | 14 | 12 | 1 | 10 | 10 | 7 | 7 | 3 | 10 | 7 | 9 | 9 | 4 | 4
  CFA/I: No | 0 | 0 | 14 | 0 | 3 | 1 | 1 | 3 | 48 | 3 | 5 | 6 | 6 | 36 | 20 | 23 | 15 | 17 | 25 | 45
  CS3: Yes | 15 | 15 | 3 | 15 | 13 | 15 | 11 | 15 | 6 | 7 | 11 | 11 | 6 | 3 | 10 | 7 | 7 | 7 | 8 | 6
  CS3: No | 0 | 0 | 11 | 0 | 2 | 0 | 4 | 0 | 43 | 6 | 4 | 2 | 7 | 36 | 20 | 23 | 17 | 19 | 21 | 43
  CS5: Yes | 15 | 15 | 0 | 14 | 13 | 12 | 11 | 9 | 1 | 6 | 7 | 5 | 8 | 1 | 8 | 2 | 3 | 3 | 2 | 3
  CS5: No | 0 | 0 | 14 | 1 | 2 | 3 | 4 | 6 | 48 | 7 | 8 | 8 | 5 | 38 | 22 | 28 | 21 | 23 | 27 | 46
  CS6: number analyzed (Participants) | 15 | 15 | 14 | 15 | 15 | 15 | 15 | 15 | 49 | 12 | 15 | 13 | 13 | 39 | 30 | 30 | 24 | 26 | 29 | 49
  CS6: Yes | 15 | 15 | 1 | 11 | 7 | 12 | 8 | 9 | 0 | 3 | 4 | 8 | 3 | 1 | 2 | 1 | 0 | 0 | 1 | 0
  CS6: No | 0 | 0 | 13 | 4 | 8 | 3 | 7 | 6 | 49 | 9 | 11 | 5 | 10 | 38 | 28 | 29 | 24 | 26 | 28 | 49
  LTB: Yes | 15 | 15 | 0 | 15 | 15 | 15 | 15 | 14 | 2 | 11 | 15 | 13 | 11 | 3 | 15 | 20 | 18 | 15 | 19 | 8
  LTB: No | 0 | 0 | 14 | 0 | 0 | 0 | 0 | 1 | 47 | 2 | 0 | 0 | 2 | 36 | 15 | 10 | 6 | 11 | 10 | 41

5. Secondary Outcome: Geometric Mean Titer (GMT) of Antibody Lymphocyte Supernatant (ALS) Immunoglobulin A (IgA) Response After Either Vaccine Dose, by Antigen
Description: as for outcome 3
Time Frame: 19 days
Population: Subjects who received both vaccinations and had valid baseline and endline immunologic samples.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Adult: ETVAX (Full) | Adult: ETVAX (Full) + 10 ug dmLT | Adult: Placebo | 24-59 Months: ETVAX (1/4) | 24-59 Months: ETVAX (1/2) | 24-59 Months: ETVAX (1/2) + 2.5 ug dmLT | 24-59 Months: ETVAX (1/2) + 5 ug dmLT | 24-59 Months: ETVAX (1/2) + 10 ug dmLT | 24-59 Months: Placebo | 12-23 Months: ETVAX (1/4) | 12-23 Months: ETVAX (1/2) | 12-23 Months: ETVAX (1/2) + 2.5 ug dmLT | 12-23 Months: ETVAX (1/2) + 5 ug dmLT | 12-23 Months: Placebo | 6-11 Months: ETVAX (1/8) | 6-11 Months: ETVAX (1/4) | 6-11 Months: ETVAX (1/2) | 6-11 Months: ETVAX (1/4) + 2.5 ug dmLT | 6-11 Month Olds: ETVAX (1/4) + 5 ug dmLT | 6-11 Month Olds: Placebo
Number analyzed (Participants) | 15 | 15 | 14 | 15 | 15 | 15 | 15 | 15 | 49 | 13 | 15 | 13 | 13 | 39 | 30 | 30 | 24 | 26 | 29 | 49
titer
  CFA/I | 9991 [5436 to 18363] | 6732 [4023 to 11264] | 115 [96.6 to 137] | 7298 [3881 to 13724] | 2913 [1051 to 8072] | 7819 [3265 to 18726] | 2239 [980 to 5114] | 3164 [1014 to 9878] | 149 [135 to 165] | 1490 [594 to 3741] | 2937 [783 to 11013] | 577 [175 to 1900] | 862 [262 to 2842] | 155 [108 to 222] | 318 [156 to 649] | 228 [108 to 480] | 328 [143 to 755] | 202 [94.7 to 429] | 123 [79.3 to 191] | 104 [78.8 to 138]
  CS3 | 11354 [6183 to 20848] | 7658 [4208 to 13937] | 221 [115 to 424] | 9277 [4408 to 19525] | 2283 [923 to 5646] | 4868 [2564 to 9243] | 1400 [639 to 3063] | 4076 [2240 to 7419] | 190 [154 to 234] | 600 [240 to 1502] | 1322 [601 to 2906] | 1346 [470 to 3853] | 700 [208 to 2360] | 134 [106 to 169] | 355 [198 to 639] | 263 [138 to 501] | 212 [122 to 368] | 186 [116 to 298] | 196 [118 to 324] | 123 [92.8 to 164]
  CS5 | 4405 [2264 to 8573] | 5198 [2647 to 10204] | 101 [87.9 to 116] | 4869 [1987 to 11930] | 1473 [689 to 3148] | 1921 [620 to 5955] | 876 [357 to 2145] | 913 [246 to 3386] | 96.3 [86.8 to 107] | 369 [140 to 973] | 394 [144 to 1076] | 229 [89.8 to 586] | 616 [200 to 1897] | 83.3 [73.9 to 94.0] | 163 [102 to 261] | 100 [71.0 to 141] | 190 [144 to 251] | 90.4 [64.8 to 126] | 81.5 [56.5 to 118] | 99.9 [83.2 to 120]
  CS6: number analyzed (Participants) | 15 | 15 | 14 | 15 | 15 | 15 | 15 | 15 | 49 | 13 | 15 | 13 | 13 | 37 | 30 | 30 | 24 | 26 | 29 | 49
  CS6 | 5535 [2947 to 10398] | 4795 [2781 to 8267] | 126 [96.5 to 164] | 727 [297 to 1783] | 440 [194 to 997] | 990 [479 to 2045] | 468 [254 to 862] | 255 [101 to 646] | 76.1 [69.0 to 83.9] | 210 [93.6 to 471] | 187 [93.3 to 374] | 225 [115 to 441] | 325 [139 to 762] | 93.9 [78.5 to 112] | 110 [92.3 to 131] | 89.6 [75.5 to 106] | 82.7 [71.8 to 95.3] | 60.9 [55.5 to 66.8] | 60.9 [55.5 to 66.8] | 96.3 [84.2 to 110]
  LTB | 3184 [2007 to 5052] | 3450 [1685 to 7065] | 82.1 [76.8 to 87.6] | 2545 [1074 to 6028] | 2067 [1190 to 3589] | 6417 [2978 to 13829] | 1435 [854 to 2411] | 2475 [1135 to 5400] | 71.5 [64.4 to 79.4] | 914 [436 to 1914] | 1883 [1106 to 3206] | 2242 [973 to 5163] | 1584 [534 to 4697] | 91.7 [77.3 to 109] | 396 [242 to 648] | 704 [387 to 1283] | 506 [299 to 856] | 771 [326 to 1823] | 509 [276 to 939] | 129 [97.7 to 171]

6. Secondary Outcome: Geometric Mean Fold Change of Antibody Lymphocyte Supernatant (ALS) Immunoglobulin A (IgA) Response After Either Vaccine Dose, by Antigen
Description: as for outcome 3
Time Frame: 19 days
Population: Subjects who received both vaccinations and had valid baseline and endline immunologic samples.
Measure: Geometric Mean (95% Confidence Interval); unit: fold change
Arm/Group | Adult: ETVAX (Full) | Adult: ETVAX (Full) + 10 ug dmLT | Adult: Placebo | 24-59 Months: ETVAX (1/4) | 24-59 Months: ETVAX (1/2) | 24-59 Months: ETVAX (1/2) + 2.5 ug dmLT | 24-59 Months: ETVAX (1/2) + 5 ug dmLT | 24-59 Months: ETVAX (1/2) + 10 ug dmLT | 24-59 Months: Placebo | 12-23 Months: ETVAX (1/4) | 12-23 Months: ETVAX (1/2) | 12-23 Months: ETVAX (1/2) + 2.5 ug dmLT | 12-23 Months: ETVAX (1/2) + 5 ug dmLT | 12-23 Months: Placebo | 6-11 Months: ETVAX (1/8) | 6-11 Months: ETVAX (1/4) | 6-11 Months: ETVAX (1/2) | 6-11 Months: ETVAX (1/4) + 2.5 ug dmLT | 6-11 Month Olds: ETVAX (1/4) + 5 ug dmLT | 6-11 Month Olds: Placebo
Number analyzed (Participants) | 15 | 15 | 14 | 15 | 15 | 15 | 15 | 15 | 49 | 13 | 15 | 13 | 13 | 39 | 30 | 30 | 24 | 26 | 29 | 49
fold change
  CFA/I | 97 [48.6 to 193] | 73.6 [46.6 to 116] | 1.11 [0.981 to 1.26] | 82.6 [44.5 to 153] | 22.5 [8.14 to 62.1] | 82.9 [33.5 to 205] | 26.9 [11.7 to 61.5] | 35.2 [11.3 to 110] | 1.43 [1.30 to 1.58] | 17.5 [6.49 to 47.3] | 31.9 [8.14 to 125] | 9.24 [2.81 to 30.4] | 11.3 [3.45 to 36.8] | 1.69 [1.19 to 2.41] | 4.26 [2.07 to 8.78] | 2.96 [1.42 to 6.16] | 4.75 [2.07 to 10.9] | 3.67 [1.72 to 7.80] | 1.81 [1.17 to 2.80] | 1.54 [1.15 to 2.06]
  CS3 | 97.5 [51.5 to 185] | 74.5 [40.8 to 136] | 1.91 [0.979 to 3.73] | 85.2 [41.0 to 177] | 16.8 [6.96 to 40.4] | 38.2 [20.3 to 71.9] | 15.3 [6.97 to 33.4] | 34 [18.7 to 61.8] | 1.6 [1.32 to 1.94] | 7.38 [2.95 to 18.5] | 13.2 [6.07 to 28.8] | 21.1 [7.38 to 60.2] | 5.83 [1.73 to 19.7] | 1.56 [1.29 to 1.89] | 3.67 [2.07 to 6.50] | 3.39 [1.78 to 6.46] | 2.95 [1.70 to 5.12] | 2.81 [1.75 to 4.52] | 2.72 [1.64 to 4.50] | 1.62 [1.23 to 2.13]
  CS5 | 44.5 [23.0 to 86.3] | 57.1 [28.5 to 114] | 1.05 [0.937 to 1.18] | 57.2 [23.2 to 141] | 20.2 [9.40 to 43.3] | 26.5 [8.44 to 82.9] | 12.3 [4.99 to 30.1] | 11.1 [2.98 to 41.0] | 1.26 [1.14 to 1.39] | 4.62 [1.68 to 12.7] | 5.26 [1.87 to 14.8] | 3.67 [1.44 to 9.37] | 8.92 [2.89 to 27.5] | 1.16 [1.02 to 1.31] | 2.52 [1.58 to 4.03] | 1.54 [1.09 to 2.17] | 1.58 [1.20 to 2.09] | 1.48 [1.06 to 2.07] | 1.29 [0.897 to 1.87] | 1.37 [1.15 to 1.62]
  CS6: number analyzed (Participants) | 15 | 15 | 14 | 15 | 15 | 15 | 15 | 15 | 49 | 13 | 15 | 13 | 13 | 37 | 30 | 30 | 24 | 26 | 29 | 49
  CS6 | 65.6 [33.8 to 127] | 59.4 [34.1 to 103] | 1.43 [1.08 to 1.89] | 12.5 [5.10 to 30.7] | 7.1 [3.14 to 16.1] | 14.9 [7.01 to 31.6] | 5.84 [3.17 to 10.8] | 6 [2.37 to 15.2] | 1.28 [1.19 to 1.37] | 3.2 [1.41 to 7.28] | 2.83 [1.36 to 5.87] | 3.98 [2.04 to 7.76] | 2.96 [1.26 to 6.93] | 1.33 [1.15 to 1.53] | 1.3 [1.11 to 1.52] | 1.38 [1.16 to 1.64] | 1.5 [1.31 to 1.73] | 1.03 [0.941 to 1.13] | 1.38 [1.20 to 1.57] | 1.24 [1.14 to 1.34]
  LTB | 45.5 [28.7 to 72.2] | 49.3 [24.1 to 101] | 1.17 [1.10 to 1.25] | 44.3 [19.5 to 101] | 36.9 [21.2 to 64.2] | 106 [49.7 to 225] | 25 [14.9 to 41.9] | 41.3 [18.9 to 90.0] | 1.23 [1.10 to 1.38] | 16 [7.65 to 33.6] | 35.6 [21.3 to 59.7] | 39 [16.9 to 89.8] | 16.2 [5.48 to 48.2] | 1.47 [1.26 to 1.71] | 4.85 [2.94 to 7.99] | 8.8 [4.83 to 16.0] | 7.55 [4.46 to 12.8] | 12.6 [5.34 to 29.9] | 9.25 [5.01 to 17.1] | 1.91 [1.45 to 2.52]

7. Secondary Outcome: Number and Percentage of 6-11 Month Old Subjects With ≥Two-fold Increase in Fecal Secretory Immunoglobulin A (SIgA) Response, by Antigen
Description: Fecal secretion was measured on Day 7, Day 19, and Day 28; number in table is subjects experiencing a two-fold rise at any of these time points. Antigen in ETVAX were:
  E. coli, CFA/I, strain ETEX 21 formalin inactivated, E. coli, CS3, strain ETEX 22 formalin inactivated, E. coli, CS5, strain ETEX 23 formalin inactivated, E. coli, CS6, strain ETEX 24 phenol inactivated, B-subunit of the E. coli heat-labile enterotoxin
Time Frame: 28 days
Population: Subjects who received both vaccinations and had valid baseline and endline immunologic samples.
Measure: Count of Participants; unit: Participants
Arm/Group | 6-11 Months: ETVAX (1/8) | 6-11 Months: ETVAX (1/4) | 6-11 Months: ETVAX (1/2) | 6-11 Months: ETVAX (1/4) + 2.5 ug dmLT | 6-11 Month Olds: ETVAX (1/4) + 5 ug dmLT | 6-11 Month Olds: Placebo
Number analyzed (Participants) | 23 | 23 | 16 | 20 | 21 | 37
Participants
  CFA/I: number analyzed (Participants) | 20 | 20 | 15 | 19 | 14 | 32
  CFA/I: Yes | 15 | 10 | 9 | 13 | 8 | 16
  CFA/I: No | 5 | 10 | 6 | 6 | 6 | 16
  CS3: number analyzed (Participants) | 21 | 22 | 16 | 20 | 18 | 35
  CS3: Yes | 12 | 10 | 9 | 14 | 14 | 19
  CS3: No | 9 | 12 | 7 | 6 | 4 | 16
  CS5: number analyzed (Participants) | 20 | 21 | 16 | 19 | 15 | 30
  CS5: Yes | 12 | 10 | 9 | 12 | 7 | 11
  CS5: No | 8 | 11 | 7 | 7 | 8 | 19
  CS6: number analyzed (Participants) | 20 | 22 | 14 | 19 | 18 | 33
  CS6: Yes | 11 | 13 | 8 | 15 | 6 | 10
  CS6: No | 9 | 9 | 6 | 4 | 12 | 23
  LTB: number analyzed (Participants) | 22 | 22 | 16 | 20 | 21 | 36
  LTB: Yes | 14 | 15 | 14 | 15 | 14 | 20
  LTB: No | 8 | 7 | 2 | 5 | 7 | 16

8. Secondary Outcome: Number and Percentage of 6-11 Month Old Subjects With ≥Four-fold Increase in Fecal Secretory Immunoglobulin A (SIgA) Response, by Antigen
Description: Fecal secretion was measured on Day 7, Day 19, and Day 28; number in table is subjects experiencing a four-fold rise at any of these time points. Antigens in ETVAX were:
  E. coli, CFA/I, strain ETEX 21 formalin inactivated, E. coli, CS3, strain ETEX 22 formalin inactivated, E. coli, CS5, strain ETEX 23 formalin inactivated, E. coli, CS6, strain ETEX 24 phenol inactivated, B-subunit of the E. coli heat-labile enterotoxin
Time Frame: 28 days
Population: Subjects who received both vaccinations and had valid baseline and endline immunologic samples.
Measure: Count of Participants; unit: Participants
Arm/Group | 6-11 Months: ETVAX (1/8) | 6-11 Months: ETVAX (1/4) | 6-11 Months: ETVAX (1/2) | 6-11 Months: ETVAX (1/4) + 2.5 ug dmLT | 6-11 Month Olds: ETVAX (1/4) + 5 ug dmLT | 6-11 Month Olds: Placebo
Number analyzed (Participants) | 23 | 23 | 16 | 20 | 21 | 37
Participants
  CFA/I: number analyzed (Participants) | 20 | 20 | 15 | 19 | 14 | 32
  CFA/I: Yes | 8 | 6 | 7 | 10 | 6 | 8
  CFA/I: No | 12 | 14 | 8 | 9 | 8 | 24
  CS3: number analyzed (Participants) | 21 | 22 | 16 | 20 | 18 | 35
  CS3: Yes | 6 | 6 | 4 | 8 | 8 | 9
  CS3: No | 15 | 16 | 12 | 12 | 10 | 26
  CS5: number analyzed (Participants) | 20 | 21 | 16 | 19 | 15 | 30
  CS5: Yes | 6 | 5 | 9 | 10 | 2 | 5
  CS5: No | 14 | 16 | 7 | 9 | 13 | 25
  CS6: number analyzed (Participants) | 20 | 22 | 14 | 19 | 18 | 33
  CS6: Yes | 5 | 7 | 5 | 12 | 3 | 9
  CS6: No | 15 | 15 | 9 | 7 | 15 | 24
  LTB: number analyzed (Participants) | 22 | 22 | 16 | 20 | 21 | 36
  LTB: Yes | 11 | 11 | 10 | 13 | 10 | 10
  LTB: No | 11 | 11 | 6 | 7 | 11 | 26

9. Secondary Outcome: Geometric Mean Titer (GMT) of Fecal Secretory Immunoglobulin A (SIgA) Response 6-11 Month Old Subjects, by Antigen
Description: Fecal secretion was measured on Day 7, Day 19, and Day 28; number in table is based on the maximum value for each subject. Antigen in ETVAX were:
  E. coli, CFA/I, strain ETEX 21 formalin inactivated, E. coli, CS3, strain ETEX 22 formalin inactivated, E. coli, CS5, strain ETEX 23 formalin inactivated, E. coli, CS6, strain ETEX 24 phenol inactivated, B-subunit of the E. coli heat-labile enterotoxin
Time Frame: 28 days
Population: Subjects who received both vaccinations and had valid baseline and endline immunologic samples.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 6-11 Months: ETVAX (1/8) | 6-11 Months: ETVAX (1/4) | 6-11 Months: ETVAX (1/2) | 6-11 Months: ETVAX (1/4) + 2.5 ug dmLT | 6-11 Month Olds: ETVAX (1/4) + 5 ug dmLT | 6-11 Month Olds: Placebo
Number analyzed (Participants) | 23 | 23 | 16 | 20 | 21 | 37
titer
  CFA/I: number analyzed (Participants) | 20 | 20 | 16 | 19 | 14 | 32
  CFA/I | 74.3 [38.2 to 145] | 281 [137 to 578] | 141 [69.5 to 285] | 230 [126 to 418] | 122 [72.6 to 207] | 113 [70.0 to 183]
  CS3: number analyzed (Participants) | 21 | 22 | 16 | 20 | 18 | 35
  CS3 | 236 [94.4 to 588] | 340 [150 to 744] | 101 [44 to 230] | 332 [199 to 551] | 402 [234 to 689] | 204 [141 to 295]
  CS5: number analyzed (Participants) | 20 | 21 | 16 | 19 | 15 | 30
  CS5 | 47.7 [28.9 to 78.7] | 153 [89.7 to 263] | 63.9 [26.3 to 155] | 107 [74.9 to 153] | 127 [65.0 to 249] | 74 [49.2 to 111]
  CS6: number analyzed (Participants) | 20 | 22 | 16 | 19 | 18 | 33
  CS6 | 122 [65.9 to 226] | 272 [152 to 488] | 90.3 [46.5 to 175] | 361 [199 to 656] | 170 [102 to 281] | 181 [114 to 287]
  LTB: number analyzed (Participants) | 22 | 22 | 16 | 20 | 21 | 36
  LTB | 655 [397 to 1079] | 2330 [1140 to 4764] | 1500 [838 to 2684] | 4159 [1995 to 8672] | 1299 [600 to 2813] | 839 [549 to 1281]

10. Secondary Outcome: Geometric Mean Fold Change of Fecal Secretory Immunoglobulin A (SIgA) Response Among 6-11 Month Old Subjects, by Antigen
Description: as for outcome 9
Time Frame: 28 days
Population: Subjects who received both vaccinations and had valid baseline and endline immunologic samples.
Measure: Geometric Mean (95% Confidence Interval); unit: fold change
Arm/Group | 6-11 Months: ETVAX (1/8) | 6-11 Months: ETVAX (1/4) | 6-11 Months: ETVAX (1/2) | 6-11 Months: ETVAX (1/4) + 2.5 ug dmLT | 6-11 Month Olds: ETVAX (1/4) + 5 ug dmLT | 6-11 Month Olds: Placebo
Number analyzed (Participants) | 23 | 23 | 16 | 20 | 21 | 37
fold change
  CFA/I: number analyzed (Participants) | 20 | 20 | 15 | 19 | 14 | 32
  CFA/I | 3.59 [2.19 to 5.90] | 3.36 [1.60 to 7.05] | 3.41 [1.31 to 8.90] | 5.19 [2.37 to 11.4] | 2.7 [1.28 to 5.73] | 2.1 [1.21 to 3.62]
  CS3: number analyzed (Participants) | 21 | 22 | 16 | 20 | 18 | 35
  CS3 | 2.98 [1.80 to 4.92] | 2.57 [1.32 to 5.00] | 2 [0.743 to 5.38] | 4.6 [2.18 to 9.74] | 3.66 [2.22 to 6.02] | 1.91 [1.28 to 2.84]
  CS5: number analyzed (Participants) | 20 | 21 | 16 | 19 | 15 | 30
  CS5 | 2.47 [1.50 to 4.07] | 2.63 [1.42 to 4.85] | 3.96 [1.41 to 11.1] | 4.08 [2.14 to 7.77] | 1.78 [1.03 to 3.06] | 1.79 [1.12 to 2.84]
  CS6: number analyzed (Participants) | 20 | 22 | 14 | 19 | 18 | 33
  CS6 | 1.76 [0.937 to 3.30] | 2.85 [1.53 to 5.31] | 1.4 [0.362 to 5.40] | 7.21 [3.44 to 15.1] | 1.72 [1.08 to 2.73] | 1.96 [1.21 to 3.18]
  LTB: number analyzed (Participants) | 22 | 22 | 16 | 20 | 21 | 36
  LTB | 3.74 [1.82 to 7.68] | 3.71 [2.01 to 6.87] | 8.3 [4.18 to 16.5] | 8.8 [3.73 to 20.8] | 5.64 [2.31 to 13.8] | 2.58 [1.52 to 4.36]

11. Secondary Outcome: Number and Percentage of Subjects With ≥Two-fold Increase in Plasma Immunoglobulin A (IgA) Response After Either Vaccine Dose, for Antigens in ETVAX
Description: as for outcome 3
Time Frame: 19 days
Population: Subjects who received both vaccinations and had valid baseline and endline immunologic samples.
Measure: Count of Participants; unit: Participants
Arm/Group | Adult: ETVAX (Full) | Adult: ETVAX (Full) + 10 ug dmLT | Adult: Placebo | 24-59 Months: ETVAX (1/4) | 24-59 Months: ETVAX (1/2) | 24-59 Months: ETVAX (1/2) + 2.5 ug dmLT | 24-59 Months: ETVAX (1/2) + 5 ug dmLT | 24-59 Months: ETVAX (1/2) + 10 ug dmLT | 24-59 Months: Placebo | 12-23 Months: ETVAX (1/4) | 12-23 Months: ETVAX (1/2) | 12-23 Months: ETVAX (1/2) + 2.5 ug dmLT | 12-23 Months: ETVAX (1/2) + 5 ug dmLT | 12-23 Months: Placebo | 6-11 Months: ETVAX (1/8) | 6-11 Months: ETVAX (1/4) | 6-11 Months: ETVAX (1/2) | 6-11 Months: ETVAX (1/4) + 2.5 ug dmLT | 6-11 Month Olds: ETVAX (1/4) + 5 ug dmLT | 6-11 Month Olds: Placebo
Number analyzed (Participants) | 15 | 15 | 14 | 15 | 15 | 15 | 15 | 15 | 49 | 13 | 15 | 13 | 13 | 39 | 30 | 30 | 25 | 26 | 29 | 49
Participants
  CFA/I: Yes | 12 | 14 | 0 | 13 | 10 | 11 | 12 | 12 | 3 | 7 | 11 | 5 | 8 | 8 | 12 | 14 | 11 | 12 | 14 | 15
  CFA/I: No | 3 | 1 | 14 | 2 | 5 | 4 | 3 | 3 | 46 | 6 | 4 | 8 | 5 | 31 | 18 | 16 | 14 | 14 | 15 | 34
  CS3: number analyzed (Participants) | 15 | 14 | 14 | 15 | 15 | 15 | 15 | 15 | 49 | 13 | 15 | 13 | 13 | 39 | 30 | 30 | 25 | 26 | 29 | 49
  CS3: Yes | 14 | 13 | 3 | 14 | 12 | 12 | 10 | 13 | 5 | 7 | 6 | 5 | 6 | 8 | 15 | 17 | 13 | 12 | 14 | 14
  CS3: No | 1 | 1 | 11 | 1 | 3 | 3 | 5 | 2 | 44 | 6 | 9 | 8 | 7 | 31 | 15 | 13 | 12 | 14 | 15 | 35
  CS5: number analyzed (Participants) | 14 | 15 | 13 | 15 | 15 | 15 | 15 | 15 | 49 | 13 | 15 | 13 | 13 | 39 | 30 | 30 | 25 | 26 | 29 | 49
  CS5: Yes | 9 | 12 | 0 | 11 | 7 | 7 | 7 | 8 | 3 | 5 | 5 | 3 | 7 | 7 | 10 | 13 | 10 | 13 | 9 | 10
  CS5: No | 5 | 3 | 13 | 4 | 8 | 8 | 8 | 7 | 46 | 8 | 10 | 10 | 6 | 32 | 20 | 17 | 15 | 13 | 20 | 39
  CS6: number analyzed (Participants) | 13 | 15 | 13 | 15 | 15 | 15 | 15 | 15 | 49 | 13 | 15 | 13 | 13 | 39 | 30 | 30 | 25 | 26 | 29 | 49
  CS6: Yes | 8 | 11 | 0 | 5 | 12 | 8 | 8 | 5 | 3 | 6 | 5 | 3 | 5 | 6 | 11 | 9 | 9 | 11 | 12 | 14
  CS6: No | 5 | 4 | 13 | 10 | 3 | 7 | 7 | 10 | 46 | 7 | 10 | 10 | 8 | 33 | 19 | 21 | 16 | 15 | 17 | 35
  LTB: Yes | 15 | 15 | 1 | 14 | 14 | 15 | 14 | 14 | 9 | 12 | 12 | 12 | 13 | 8 | 22 | 26 | 21 | 21 | 24 | 21
  LTB: No | 0 | 0 | 13 | 1 | 1 | 0 | 1 | 1 | 40 | 1 | 3 | 1 | 0 | 31 | 8 | 4 | 4 | 5 | 5 | 28

12. Secondary Outcome: Number and Percentage of Subjects With ≥Four-fold Increase in Plasma Immunoglobulin A (IgA) Response After Either Vaccine Dose, for Antigens in ETVAX
Description: as for outcome 3
Time Frame: 19 days
Population: Subjects who received both vaccinations and had valid baseline and endline immunologic samples.
Measure: Count of Participants; unit: Participants
Arm/Group | Adult: ETVAX (Full) | Adult: ETVAX (Full) + 10 ug dmLT | Adult: Placebo | 24-59 Months: ETVAX (1/4) | 24-59 Months: ETVAX (1/2) | 24-59 Months: ETVAX (1/2) + 2.5 ug dmLT | 24-59 Months: ETVAX (1/2) + 5 ug dmLT | 24-59 Months: ETVAX (1/2) + 10 ug dmLT | 24-59 Months: Placebo | 12-23 Months: ETVAX (1/4) | 12-23 Months: ETVAX (1/2) | 12-23 Months: ETVAX (1/2) + 2.5 ug dmLT | 12-23 Months: ETVAX (1/2) + 5 ug dmLT | 12-23 Months: Placebo | 6-11 Months: ETVAX (1/8) | 6-11 Months: ETVAX (1/4) | 6-11 Months: ETVAX (1/2) | 6-11 Months: ETVAX (1/4) + 2.5 ug dmLT | 6-11 Month Olds: ETVAX (1/4) + 5 ug dmLT | 6-11 Month Olds: Placebo
Number analyzed (Participants) | 15 | 15 | 14 | 15 | 15 | 15 | 15 | 15 | 49 | 13 | 15 | 13 | 13 | 39 | 30 | 30 | 25 | 26 | 29 | 49
Participants
  CFA/I: Yes | 7 | 6 | 0 | 4 | 5 | 5 | 10 | 11 | 2 | 3 | 4 | 3 | 4 | 4 | 9 | 9 | 6 | 9 | 7 | 10
  CFA/I: No | 8 | 9 | 14 | 11 | 10 | 10 | 5 | 4 | 47 | 10 | 11 | 10 | 9 | 35 | 21 | 21 | 19 | 17 | 22 | 39
  CS3: number analyzed (Participants) | 15 | 14 | 14 | 15 | 15 | 15 | 15 | 15 | 49 | 13 | 15 | 13 | 13 | 39 | 30 | 30 | 25 | 26 | 29 | 49
  CS3: Yes | 11 | 10 | 2 | 12 | 8 | 6 | 3 | 7 | 1 | 5 | 3 | 4 | 4 | 4 | 8 | 10 | 7 | 5 | 10 | 5
  CS3: No | 4 | 4 | 12 | 3 | 7 | 9 | 12 | 8 | 48 | 8 | 12 | 9 | 9 | 35 | 22 | 20 | 18 | 21 | 19 | 44
  CS5: number analyzed (Participants) | 14 | 14 | 13 | 15 | 15 | 15 | 15 | 15 | 49 | 13 | 15 | 13 | 13 | 39 | 30 | 30 | 25 | 26 | 29 | 49
  CS5: Yes | 6 | 6 | 0 | 6 | 6 | 3 | 0 | 4 | 0 | 2 | 3 | 2 | 2 | 2 | 3 | 8 | 5 | 7 | 6 | 5
  CS5: No | 8 | 8 | 13 | 9 | 9 | 12 | 15 | 11 | 49 | 11 | 12 | 11 | 11 | 37 | 27 | 22 | 20 | 19 | 23 | 44
  CS6: number analyzed (Participants) | 13 | 15 | 13 | 15 | 15 | 15 | 15 | 15 | 49 | 13 | 15 | 13 | 13 | 39 | 30 | 30 | 25 | 26 | 29 | 49
  CS6: Yes | 4 | 5 | 0 | 3 | 6 | 4 | 2 | 2 | 1 | 3 | 1 | 1 | 3 | 4 | 4 | 2 | 4 | 7 | 5 | 7
  CS6: No | 9 | 10 | 13 | 12 | 9 | 11 | 13 | 13 | 48 | 10 | 14 | 12 | 10 | 35 | 26 | 28 | 21 | 19 | 24 | 42
  LTB: Yes | 13 | 14 | 0 | 11 | 14 | 14 | 12 | 14 | 6 | 9 | 11 | 10 | 13 | 4 | 17 | 21 | 17 | 18 | 22 | 13
  LTB: No | 2 | 1 | 14 | 4 | 1 | 1 | 3 | 1 | 43 | 4 | 4 | 3 | 0 | 35 | 13 | 9 | 8 | 8 | 7 | 36

13. Secondary Outcome: Geometric Mean Titer (GMT) of Plasma Immunoglobulin A (IgA) Response After Either Vaccine Dose, for Antigens in ETVAX
Description: as for outcome 3
Time Frame: 19 days
Population: Subjects who received both vaccinations and had valid baseline and endline immunologic samples.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Adult: ETVAX (Full) | Adult: ETVAX (Full) + 10 ug dmLT | Adult: Placebo | 24-59 Months: ETVAX (1/4) | 24-59 Months: ETVAX (1/2) | 24-59 Months: ETVAX (1/2) + 2.5 ug dmLT | 24-59 Months: ETVAX (1/2) + 5 ug dmLT | 24-59 Months: ETVAX (1/2) + 10 ug dmLT | 24-59 Months: Placebo | 12-23 Months: ETVAX (1/4) | 12-23 Months: ETVAX (1/2) | 12-23 Months: ETVAX (1/2) + 2.5 ug dmLT | 12-23 Months: ETVAX (1/2) + 5 ug dmLT | 12-23 Months: Placebo | 6-11 Months: ETVAX (1/8) | 6-11 Months: ETVAX (1/4) | 6-11 Months: ETVAX (1/2) | 6-11 Months: ETVAX (1/4) + 2.5 ug dmLT | 6-11 Month Olds: ETVAX (1/4) + 5 ug dmLT | 6-11 Month Olds: Placebo
Number analyzed (Participants) | 15 | 15 | 14 | 15 | 15 | 15 | 15 | 15 | 49 | 13 | 15 | 13 | 13 | 39 | 30 | 30 | 25 | 26 | 29 | 49
titer
  CFA/I | 74.4 [48.9 to 113] | 57.8 [39.6 to 94.4] | 20 [17.4 to 23.0] | 665 [392 to 1127] | 692 [414 to 1158] | 1036 [569 to 1887] | 669 [330 to 1356] | 677 [269 to 1705] | 265 [223 to 315] | 368 [148 to 919] | 532 [224 to 1263] | 163 [80.1 to 334] | 189 [72.0 to 496] | 115 [81.9 to 162] | 111 [64 to 192] | 133 [66.3 to 267] | 164 [83.3 to 322] | 63.4 [28.8 to 140] | 98.4 [65.8 to 147] | 59.2 [43.2 to 81.3]
  CS3 | 243 [162 to 363] | 229 [153 to 344] | 53.1 [31.1 to 90.6] | 991 [684 to 1437] | 529 [222 to 1260] | 475 [315 to 718] | 483 [309 to 754] | 1299 [752 to 2244] | 237 [189 to 297] | 318 [132 to 768] | 590 [384 to 907] | 245 [115 to 526] | 260 [103 to 656] | 141 [100 to 197] | 105 [61.2 to 181] | 140 [80.8 to 242] | 77.6 [46.5 to 130] | 45.1 [30.1 to 67.6] | 111 [74.0 to 167] | 53.8 [39.9 to 72.7]
  CS5: number analyzed (Participants) | 14 | 15 | 13 | 15 | 15 | 15 | 15 | 15 | 49 | 13 | 15 | 13 | 13 | 39 | 30 | 30 | 25 | 26 | 29 | 49
  CS5 | 35.3 [21.7 to 57.4] | 42.1 [28.9 to 61.3] | 13.6 [9.92 to 18.7] | 147 [87.9 to 247] | 131 [65.2 to 263] | 402 [290 to 558] | 317 [225 to 447] | 194 [111 to 339] | 123 [91.7 to 166] | 76.1 [37.2 to 156] | 191 [132 to 277] | 298 [219 to 405] | 203 [136 to 305] | 96.6 [67.3 to 139] | 67.3 [46.4 to 97.6] | 78.9 [53.3 to 117] | 67 [43.6 to 103] | 57.2 [37.4 to 87.5] | 129 [94.7 to 176] | 58.9 [43.5 to 79.8]
  CS6: number analyzed (Participants) | 13 | 15 | 13 | 15 | 15 | 15 | 15 | 15 | 49 | 13 | 15 | 13 | 13 | 39 | 30 | 30 | 25 | 26 | 29 | 49
  CS6 | 84.8 [55.9 to 129] | 72.1 [42.1 to 123] | 20.7 [14.4 to 29.8] | 531 [304 to 926] | 694 [416 to 1157] | 508 [286 to 904] | 424 [253 to 713] | 450 [272 to 747] | 371 [304 to 453] | 430 [241 to 770] | 269 [163 to 444] | 230 [144 to 369] | 297 [156 to 565] | 231 [162 to 328] | 110 [81.2 to 150] | 137 [91.5 to 206] | 162 [115 to 228] | 74 [46.6 to 118] | 124 [98.0 to 156] | 93.8 [71.7 to 123]
  LTB | 277 [190 to 404] | 390 [180 to 842] | 10.1 [6.01 to 16.9] | 791 [455 to 1374] | 940 [515 to 1715] | 568 [364 to 887] | 386 [209 to 715] | 469 [260 to 847] | 67.3 [50.0 to 90.6] | 518 [188 to 1425] | 352 [260 to 476] | 915 [458 to 1830] | 1439 [882 to 2347] | 89.3 [66.0 to 121] | 253 [131 to 489] | 1165 [699 to 1941] | 723 [390 to 1342] | 442 [199 to 983] | 403 [195 to 834] | 90.8 [58.9 to 140]

14. Secondary Outcome: Geometric Mean Fold Change in Plasma Immunoglobulin A (IgA) Response After Either Vaccine Dose, for Antigens in ETVAX
Description: as for outcome 3
Time Frame: 19 days
Population: Subjects who received both vaccinations and had valid baseline and endline immunologic samples.
Measure: Geometric Mean (95% Confidence Interval); unit: fold change
Arm/Group | Adult: ETVAX (Full) | Adult: ETVAX (Full) + 10 ug dmLT | Adult: Placebo | 24-59 Months: ETVAX (1/4) | 24-59 Months: ETVAX (1/2) | 24-59 Months: ETVAX (1/2) + 2.5 ug dmLT | 24-59 Months: ETVAX (1/2) + 5 ug dmLT | 24-59 Months: ETVAX (1/2) + 10 ug dmLT | 24-59 Months: Placebo | 12-23 Months: ETVAX (1/4) | 12-23 Months: ETVAX (1/2) | 12-23 Months: ETVAX (1/2) + 2.5 ug dmLT | 12-23 Months: ETVAX (1/2) + 5 ug dmLT | 12-23 Months: Placebo | 6-11 Months: ETVAX (1/8) | 6-11 Months: ETVAX (1/4) | 6-11 Months: ETVAX (1/2) | 6-11 Months: ETVAX (1/4) + 2.5 ug dmLT | 6-11 Month Olds: ETVAX (1/4) + 5 ug dmLT | 6-11 Month Olds: Placebo
Number analyzed (Participants) | 15 | 15 | 14 | 15 | 15 | 15 | 15 | 15 | 49 | 13 | 15 | 13 | 13 | 39 | 30 | 30 | 25 | 26 | 29 | 49
fold change
  CFA/I | 3.34 [2.34 to 4.77] | 3.46 [2.44 to 4.90] | 1.2 [1.06 to 1.36] | 2.92 [2.01 to 4.25] | 3.52 [2.28 to 5.44] | 3.21 [1.87 to 5.50] | 5.65 [3.02 to 10.6] | 6.84 [2.69 to 17.4] | 1.19 [1.04 to 1.37] | 2.4 [1.47 to 3.92] | 2.59 [1.49 to 4.51] | 1.68 [0.741 to 3.80] | 2.94 [1.60 to 5.41] | 1.28 [0.992 to 1.65] | 2.02 [1.30 to 3.15] | 2.2 [1.43 to 3.40] | 1.96 [1.27 to 3.02] | 3.08 [1.59 to 6.00] | 1.81 [1.30 to 2.53] | 1.62 [1.25 to 2.10]
  CS3 | 8.54 [4.72 to 15.5] | 7.43 [4.09 to 13.5] | 1.62 [1.16 to 2.25] | 5.42 [3.94 to 7.46] | 6 [2.82 to 12.8] | 3.87 [2.44 to 6.13] | 3.16 [1.79 to 5.56] | 4.3 [2.34 to 7.90] | 1.17 [1.00 to 1.36] | 2.56 [1.07 to 6.09] | 1.96 [1.30 to 2.98] | 2.15 [0.881 to 5.26] | 2.82 [1.21 to 6.60] | 1.25 [0.937 to 1.66] | 2.33 [1.57 to 3.47] | 2.54 [1.70 to 3.78] | 2.24 [1.52 to 3.31] | 2.06 [1.46 to 2.93] | 2.93 [1.80 to 4.77] | 1.53 [1.20 to 1.95]
  CS5: number analyzed (Participants) | 14 | 15 | 13 | 15 | 15 | 15 | 15 | 15 | 49 | 13 | 15 | 13 | 13 | 39 | 30 | 30 | 25 | 26 | 29 | 49
  CS5 | 2.75 [1.80 to 4.21] | 3.11 [2.20 to 4.41] | 1.03 [0.759 to 1.39] | 2.81 [1.87 to 4.24] | 3.11 [1.73 to 5.60] | 2.21 [1.48 to 3.31] | 1.62 [1.18 to 2.23] | 2.38 [1.29 to 4.37] | 1.12 [0.981 to 1.28] | 1.37 [0.650 to 2.87] | 1.73 [1.08 to 2.76] | 1.51 [0.999 to 2.28] | 2.28 [1.37 to 3.81] | 1.25 [0.967 to 1.60] | 1.54 [1.11 to 2.14] | 1.73 [1.21 to 2.48] | 1.55 [0.989 to 2.44] | 2.4 [1.55 to 3.72] | 1.83 [1.40 to 2.40] | 1.47 [1.15 to 1.88]
  CS6: number analyzed (Participants) | 13 | 15 | 13 | 15 | 15 | 15 | 15 | 15 | 49 | 13 | 15 | 13 | 13 | 39 | 30 | 30 | 25 | 26 | 29 | 49
  CS6 | 2.98 [1.55 to 5.73] | 3.57 [2.20 to 5.81] | 1.23 [1.10 to 1.37] | 1.87 [1.13 to 3.09] | 3.12 [2.24 to 4.34] | 2.93 [1.80 to 4.77] | 1.92 [1.35 to 2.74] | 1.77 [1.18 to 2.65] | 1.23 [1.06 to 1.42] | 2.02 [1.25 to 3.29] | 1.62 [1.14 to 2.30] | 1.44 [1.04 to 2.00] | 2.17 [1.38 to 3.42] | 1.28 [0.898 to 1.84] | 1.5 [1.06 to 2.10] | 1.43 [1.08 to 1.91] | 1.66 [1.22 to 2.26] | 2.08 [1.37 to 3.16] | 1.84 [1.38 to 2.43] | 1.51 [1.20 to 1.90]
  LTB | 20 [9.70 to 41.1] | 36 [14.9 to 87.1] | 0.994 [0.789 to 1.25] | 6.49 [4.00 to 10.5] | 20.2 [11.5 to 35.4] | 12.7 [8.59 to 18.8] | 9.6 [5.02 to 18.4] | 15.3 [7.22 to 32.6] | 1.41 [1.08 to 1.85] | 10.7 [3.90 to 29.4] | 5.68 [2.62 to 12.3] | 9.43 [4.32 to 20.6] | 34.8 [20.3 to 59.5] | 1.12 [0.811 to 1.53] | 5.66 [3.18 to 10.1] | 9.09 [5.28 to 15.7] | 11.6 [5.69 to 23.6] | 10.8 [5.95 to 19.6] | 13 [6.65 to 25.5] | 2.14 [1.51 to 3.04]

15. Secondary Outcome: Number and Percentage of Adult Subjects With ≥Two-fold and ≥Four-fold Increase in Plasma Immunoglobulin A (IgA) Response After Either Vaccine Dose, for O78 Antigen
Description: Between baseline and post-immunization (measured 7 days after the first dose and 5 days after the second).
Time Frame: 19 days
Population: Subjects who received both vaccinations and had valid baseline and endline immunologic samples.
Measure: Count of Participants; unit: Participants
Arm/Group | Adult: ETVAX (Full) | Adult: ETVAX (Full) + 10 ug dmLT | Adult: Placebo
Number analyzed (Participants) | 15 | 15 | 14
Participants
  ≥Two-fold: Yes | 11 | 10 | 1
  ≥Two-fold: No | 4 | 5 | 13
  ≥Four-fold: Yes | 5 | 8 | 1
  ≥Four-fold: No | 10 | 7 | 13

16. Secondary Outcome: Geometric Mean Titer (GMT) for Plasma Immunoglobulin A (IgA) Response After Either Vaccine Dose, for O78 Antigen, Among Adults
Description: Between baseline and post-immunization (measured 7 days after the first dose and 5 days after the second).
Time Frame: 19 days
Population: Subjects who received both vaccinations and had valid baseline and endline immunologic samples.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Adult: ETVAX (Full) | Adult: ETVAX (Full) + 10 ug dmLT | Adult: Placebo
Number analyzed (Participants) | 15 | 15 | 14
titer | 177 [109 to 287] | 166 [92.0 to 301] | 30.9 [17.2 to 55.7]

17. Secondary Outcome: Geometric Mean Fold Change in Plasma Immunoglobulin A (IgA) Response After Either Vaccine Dose, for O78 Antigen, Among Adults
Description: Between baseline and post-immunization (measured 7 days after the first dose and 5 days after the second).
Time Frame: 19 days
Population: Subjects who received both vaccinations and had valid baseline and endline immunologic samples.
Measure: Geometric Mean (95% Confidence Interval); unit: fold change
Arm/Group | Adult: ETVAX (Full) | Adult: ETVAX (Full) + 10 ug dmLT | Adult: Placebo
Number analyzed (Participants) | 15 | 15 | 15
fold change | 3.15 [2.27 to 4.37] | 4.66 [2.21 to 9.84] | 0.976 [0.609 to 1.56]

18. Secondary Outcome: Number and Percentage of Subjects With ≥Two-fold and ≥Four-fold Increase in Plasma Immunoglobulin G (IgG) Response to E. Coli Heat-labile Enterotoxin (LTB) After Either Vaccine Dose
Description: Between baseline and post-immunization (measured 7 days after the first dose and 5 days after the second). B-subunit of the E. coli heat-labile enterotoxin (LTB) was one of the antigens in the ETVAX vaccine.
Time Frame: 19 days
Population: Subjects who received both vaccinations and had valid baseline and endline immunologic samples.
Measure: Count of Participants; unit: Participants
Arm/Group | Adult: ETVAX (Full) | Adult: ETVAX (Full) + 10 ug dmLT | Adult: Placebo | 24-59 Months: ETVAX (1/4) | 24-59 Months: ETVAX (1/2) | 24-59 Months: ETVAX (1/2) + 2.5 ug dmLT | 24-59 Months: ETVAX (1/2) + 5 ug dmLT | 24-59 Months: ETVAX (1/2) + 10 ug dmLT | 24-59 Months: Placebo | 12-23 Months: ETVAX (1/4) | 12-23 Months: ETVAX (1/2) | 12-23 Months: ETVAX (1/2) + 2.5 ug dmLT | 12-23 Months: ETVAX (1/2) + 5 ug dmLT | 12-23 Months: Placebo | 6-11 Months: ETVAX (1/8) | 6-11 Months: ETVAX (1/4) | 6-11 Months: ETVAX (1/2) | 6-11 Months: ETVAX (1/4) + 2.5 ug dmLT | 6-11 Month Olds: ETVAX (1/4) + 5 ug dmLT | 6-11 Month Olds: Placebo
Number analyzed (Participants) | 15 | 15 | 14 | 15 | 15 | 15 | 15 | 15 | 49 | 13 | 15 | 13 | 13 | 39 | 30 | 30 | 25 | 26 | 29 | 49
Participants
  ≥Two-fold: Yes | 14 | 13 | 2 | 11 | 14 | 15 | 12 | 15 | 5 | 8 | 8 | 13 | 13 | 1 | 19 | 24 | 21 | 19 | 23 | 13
  ≥Two-fold: No | 1 | 2 | 12 | 4 | 1 | 0 | 3 | 0 | 44 | 5 | 7 | 0 | 0 | 38 | 11 | 6 | 4 | 7 | 6 | 36
  ≥Four-fold: Yes | 11 | 13 | 0 | 6 | 10 | 11 | 9 | 8 | 2 | 3 | 3 | 6 | 10 | 0 | 14 | 15 | 16 | 12 | 13 | 7
  ≥Four-fold: No | 4 | 2 | 14 | 9 | 5 | 4 | 6 | 7 | 47 | 10 | 12 | 7 | 3 | 39 | 16 | 15 | 9 | 14 | 16 | 42

19. Secondary Outcome: Geometric Mean Titer (GMT) of Plasma Immunoglobulin G (IgG) Response to E. Coli Heat-labile Enterotoxin (LTB) After Either Vaccine Dose
Description: Measured 7 days after the first dose and 5 days after the second). B-subunit of the E. coli heat-labile enterotoxin (LTB) was one of the antigens in the ETVAX vaccine.
Time Frame: 19 days
Population: Subjects who received both vaccinations and had valid baseline and endline immunologic samples.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Adult: ETVAX (Full) | Adult: ETVAX (Full) + 10 ug dmLT | Adult: Placebo | 24-59 Months: ETVAX (1/4) | 24-59 Months: ETVAX (1/2) | 24-59 Months: ETVAX (1/2) + 2.5 ug dmLT | 24-59 Months: ETVAX (1/2) + 5 ug dmLT | 24-59 Months: ETVAX (1/2) + 10 ug dmLT | 24-59 Months: Placebo | 12-23 Months: ETVAX (1/4) | 12-23 Months: ETVAX (1/2) | 12-23 Months: ETVAX (1/2) + 2.5 ug dmLT | 12-23 Months: ETVAX (1/2) + 5 ug dmLT | 12-23 Months: Placebo | 6-11 Months: ETVAX (1/8) | 6-11 Months: ETVAX (1/4) | 6-11 Months: ETVAX (1/2) | 6-11 Months: ETVAX (1/4) + 2.5 ug dmLT | 6-11 Month Olds: ETVAX (1/4) + 5 ug dmLT | 6-11 Month Olds: Placebo
Number analyzed (Participants) | 15 | 15 | 14 | 15 | 15 | 15 | 15 | 15 | 49 | 13 | 15 | 13 | 13 | 39 | 30 | 30 | 25 | 26 | 29 | 49
titer | 1582 [989 to 2530] | 1125 [589 to 2148] | 85.1 [41.2 to 176] | 5700 [3337 to 9736] | 5047 [2475 to 10291] | 3784 [2074 to 6902] | 3006 [1708 to 5290] | 2470 [1459 to 4179] | 721 [575 to 904] | 3644 [1798 to 7387] | 2401 [1539 to 3746] | 1565 [1060 to 2312] | 5163 [3144 to 8478] | 788 [636 to 976] | 1314 [747 to 2311] | 3561 [2062 to 6149] | 3935 [2522 to 6141] | 1488 [710 to 3120] | 1521 [779 to 2970] | 513 [341 to 772]

20. Secondary Outcome: Geometric Mean Fold Change of Plasma Immunoglobulin G (IgG) Response to E. Coli Heat-labile Enterotoxin (LTB) After Either Vaccine Dose
Description: Between baseline and after vaccination (measured 7 days after the first dose and 5 days after the second). B-subunit of the E. coli heat-labile enterotoxin (LTB) was one of the antigens in the ETVAX vaccine.
Time Frame: 19 days
Population: Subjects who received both vaccinations and had valid baseline and endline immunologic samples.
Measure: Geometric Mean (95% Confidence Interval); unit: fold change
Arm/Group | Adult: ETVAX (Full) | Adult: ETVAX (Full) + 10 ug dmLT | Adult: Placebo | 24-59 Months: ETVAX (1/4) | 24-59 Months: ETVAX (1/2) | 24-59 Months: ETVAX (1/2) + 2.5 ug dmLT | 24-59 Months: ETVAX (1/2) + 5 ug dmLT | 24-59 Months: ETVAX (1/2) + 10 ug dmLT | 24-59 Months: Placebo | 12-23 Months: ETVAX (1/4) | 12-23 Months: ETVAX (1/2) | 12-23 Months: ETVAX (1/2) + 2.5 ug dmLT | 12-23 Months: ETVAX (1/2) + 5 ug dmLT | 12-23 Months: Placebo | 6-11 Months: ETVAX (1/8) | 6-11 Months: ETVAX (1/4) | 6-11 Months: ETVAX (1/2) | 6-11 Months: ETVAX (1/4) + 2.5 ug dmLT | 6-11 Month Olds: ETVAX (1/4) + 5 ug dmLT | 6-11 Month Olds: Placebo
Number analyzed (Participants) | 15 | 15 | 14 | 15 | 15 | 15 | 15 | 15 | 49 | 13 | 15 | 13 | 13 | 39 | 30 | 30 | 25 | 26 | 29 | 49
fold change | 6.53 [3.92 to 10.9] | 10.3 [5.69 to 18.6] | 1.11 [0.807 to 1.53] | 3.53 [2.26 to 5.49] | 7.57 [4.47 to 12.8] | 6.39 [3.83 to 10.7] | 5.02 [3.16 to 7.98] | 4.69 [3.16 to 7.98] | 1.23 [1.05 to 1.43] | 3.56 [1.60 to 7.91] | 2.21 [1.63 to 3.01] | 4.73 [3.18 to 7.04] | 8.77 [5.35 to 14.4] | 0.996 [0.893 to 1.11] | 4.3 [2.71 to 6.81] | 5.64 [3.52 to 9.04] | 5.47 [3.42 to 8.73] | 5.19 [2.97 to 9.05] | 5.67 [3.29 to 9.77] | 1.74 [1.37 to 2.22]

21. Secondary Outcome: Number of Antigen Responses in Antibody Lymphocyte Supernatant (ALS) Immunoglobulin A (IgA) Experienced by Subjects
Time Frame: 19 days
Measure: Count of Participants; unit: Participants
Arm/Group | Adult: Placebo | Adult: ETVAX (Full) | Adult: ETVAX (Full) + 10 ug dmLT | 24-59 Months: Placebo | 24-59 Months: ETVAX (1/4) | 24-59 Months: ETVAX (1/2) | 24-59 Months: ETVAX (1/2) + 2.5 ug dmLT | 24-59 Months: ETVAX (1/2) + 5 ug dmLT | 24-59 Months: ETVAX (1/2) + 10 ug dmLT | 12-23 Months: Placebo | 12-23 Months: ETVAX (1/4) | 12-23 Months: ETVAX (1/2) | 12-23 Months: ETVAX (1/2) + 2.5 ug dmLT | 12-23 Months: ETVAX (1/2) + 5 ug dmLT | 6-11 Month Olds: Placebo | 6-11 Months: ETVAX (1/8) | 6-11 Months: ETVAX (1/4) | 6-11 Months: ETVAX (1/2) | 6-11 Months: ETVAX (1/4) + 2.5 ug dmLT | 6-11 Month Olds: ETVAX (1/4) + 5 ug dmLT
Number analyzed (Participants) | 14 | 15 | 15 | 49 | 15 | 15 | 15 | 15 | 15 | 37 | 12 | 15 | 13 | 13 | 49 | 30 | 30 | 24 | 26 | 29
Participants
  ≥Two-fold: 5 antigens | 0 | 15 | 15 | 0 | 12 | 9 | 11 | 10 | 7 | 0 | 5 | 4 | 5 | 2 | 0 | 2 | 2 | 1 | 0 | 0
  ≥Two-fold: 4 antigens | 0 | 0 | 0 | 1 | 2 | 5 | 4 | 3 | 5 | 2 | 3 | 3 | 2 | 6 | 1 | 5 | 0 | 3 | 2 | 2
  ≥Two-fold: 3 antigens | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 1 | 1 | 5 | 4 | 1 | 1 | 5 | 7 | 5 | 7 | 4
  ≥Two-fold: 2 antigens | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 2 | 0 | 3 | 3 | 1 | 2 | 1 | 7 | 7 | 8 | 10 | 4 | 6
  ≥Two-fold: 1 antigen | 5 | 0 | 0 | 9 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 2 | 0 | 1 | 18 | 4 | 10 | 3 | 9 | 13
  ≥Two-fold: 0 antigens | 9 | 0 | 0 | 37 | 0 | 0 | 0 | 0 | 0 | 26 | 0 | 0 | 0 | 2 | 22 | 7 | 3 | 2 | 4 | 4
  ≥Four-fold: 5 antigens | 0 | 15 | 15 | 0 | 11 | 4 | 10 | 5 | 5 | 0 | 1 | 3 | 3 | 2 | 0 | 1 | 0 | 0 | 0 | 0
  ≥Four-fold: 4 antigens | 0 | 0 | 0 | 0 | 3 | 9 | 4 | 6 | 5 | 0 | 3 | 3 | 3 | 2 | 1 | 2 | 1 | 0 | 0 | 0
  ≥Four-fold: 3 antigens | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 4 | 0 | 4 | 4 | 4 | 5 | 0 | 6 | 3 | 5 | 5 | 2
  ≥Four-fold: 2 antigens | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 1 | 3 | 2 | 3 | 2 | 0 | 2 | 4 | 4 | 6 | 5 | 7
  ≥Four-fold: 1 antigen | 4 | 0 | 0 | 7 | 0 | 0 | 0 | 0 | 0 | 4 | 2 | 2 | 1 | 2 | 13 | 6 | 16 | 10 | 9 | 14
  ≥Four-fold: 0 antigens | 10 | 0 | 0 | 41 | 0 | 0 | 0 | 0 | 0 | 30 | 0 | 0 | 0 | 2 | 33 | 11 | 6 | 3 | 7 | 6

22. Secondary Outcome: Number of Antigen Responses in Plasma Immunoglobulin A (IgA) Experienced by Subjects
Time Frame: 19 days
Population: Participants with results for all antigens (CFA/I, CS3, CS5, CS6, LTB) tested for.
Measure: Count of Participants; unit: Participants
Arm/Group | Adult: Placebo | Adult: ETVAX (Full) | Adult: ETVAX (Full) + 10 ug dmLT | 24-59 Months: Placebo | 24-59 Months: ETVAX (1/4) | 24-59 Months: ETVAX (1/2) | 24-59 Months: ETVAX (1/2) + 2.5 ug dmLT | 24-59 Months: ETVAX (1/2) + 5 ug dmLT | 24-59 Months: ETVAX (1/2) + 10 ug dmLT | 12-23 Months: Placebo | 12-23 Months: ETVAX (1/4) | 12-23 Months: ETVAX (1/2) | 12-23 Months: ETVAX (1/2) + 2.5 ug dmLT | 12-23 Months: ETVAX (1/2) + 5 ug dmLT | 6-11 Month Olds: Placebo | 6-11 Months: ETVAX (1/8) | 6-11 Months: ETVAX (1/4) | 6-11 Months: ETVAX (1/2) | 6-11 Months: ETVAX (1/4) + 2.5 ug dmLT | 6-11 Month Olds: ETVAX (1/4) + 5 ug dmLT
Number analyzed (Participants) | 13 | 13 | 14 | 49 | 15 | 15 | 15 | 15 | 15 | 39 | 13 | 15 | 13 | 13 | 49 | 30 | 30 | 25 | 26 | 29
Participants
  ≥Two-fold: 5 antigens | 0 | 5 | 8 | 1 | 4 | 5 | 5 | 3 | 3 | 2 | 2 | 2 | 1 | 4 | 4 | 5 | 6 | 6 | 9 | 7
  ≥Two-fold: 4 antigens | 0 | 4 | 5 | 0 | 6 | 3 | 2 | 6 | 3 | 2 | 2 | 3 | 1 | 2 | 4 | 6 | 2 | 2 | 1 | 2
  ≥Two-fold: 3 antigens | 0 | 3 | 0 | 1 | 4 | 5 | 5 | 3 | 7 | 2 | 3 | 2 | 3 | 1 | 5 | 2 | 8 | 2 | 0 | 5
  ≥Two-fold: 2 antigens | 1 | 0 | 0 | 4 | 0 | 1 | 2 | 1 | 2 | 2 | 4 | 4 | 3 | 2 | 7 | 4 | 5 | 6 | 8 | 3
  ≥Two-fold: 1 antigen | 2 | 1 | 1 | 7 | 1 | 1 | 1 | 1 | 0 | 9 | 2 | 3 | 4 | 4 | 9 | 7 | 7 | 8 | 4 | 9
  ≥Two-fold: 0 antigens | 10 | 0 | 0 | 36 | 0 | 0 | 0 | 1 | 0 | 22 | 0 | 1 | 1 | 0 | 20 | 6 | 2 | 1 | 4 | 3
  ≥Four-fold: 5 antigens | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 1 | 2 | 3 | 3
  ≥Four-fold: 4 antigens | 0 | 4 | 2 | 0 | 0 | 4 | 2 | 0 | 1 | 2 | 2 | 2 | 1 | 1 | 2 | 1 | 2 | 0 | 1 | 2
  ≥Four-fold: 3 antigens | 0 | 2 | 4 | 1 | 4 | 5 | 2 | 4 | 5 | 2 | 1 | 1 | 0 | 2 | 2 | 2 | 5 | 2 | 4 | 2
  ≥Four-fold: 2 antigens | 0 | 1 | 6 | 2 | 9 | 2 | 3 | 5 | 6 | 0 | 4 | 2 | 3 | 2 | 5 | 5 | 7 | 5 | 5 | 3
  ≥Four-fold: 1 antigen | 2 | 5 | 0 | 3 | 1 | 4 | 7 | 5 | 2 | 4 | 3 | 7 | 5 | 7 | 11 | 11 | 8 | 13 | 5 | 15
  ≥Four-fold: 0 antigens | 11 | 0 | 1 | 43 | 0 | 0 | 0 | 1 | 0 | 31 | 3 | 3 | 3 | 0 | 28 | 9 | 7 | 3 | 8 | 4

23. Secondary Outcome: Number and Percentage of 6-11 Month Old Subjects With ≥Two-fold Increase in Fecal Secretory Immunoglobulin A (SIgA) Response on Day 7, by Antigen
Description: Fecal secretion was measured on Day 0 and Day 7 (7 days after administration of first dose of vaccine). Antigens in ETVAX were:
  E. coli, CFA/I, strain ETEX 21 formalin inactivated, E. coli, CS3, strain ETEX 22 formalin inactivated, E. coli, CS5, strain ETEX 23 formalin inactivated, E. coli, CS6, strain ETEX 24 phenol inactivated, B-subunit of the E. coli heat-labile enterotoxin
Time Frame: 7 days
Population: Subjects who received both vaccinations and had valid baseline and endline immunologic samples.
Measure: Count of Participants; unit: Participants
Arm/Group | 6-11 Months: ETVAX (1/8) | 6-11 Months: ETVAX (1/4) | 6-11 Months: ETVAX (1/2) | 6-11 Months: ETVAX (1/4) + 2.5 ug dmLT | 6-11 Month Olds: ETVAX (1/4) + 5 ug dmLT | 6-11 Month Olds: Placebo
Number analyzed (Participants) | 23 | 23 | 16 | 20 | 21 | 37
Participants
  CFA/I: number analyzed (Participants) | 16 | 13 | 11 | 16 | 13 | 21
  CFA/I: Yes | 8 | 2 | 3 | 10 | 7 | 6
  CFA/I: No | 8 | 11 | 8 | 6 | 6 | 15
  CS3: number analyzed (Participants) | 17 | 15 | 12 | 17 | 16 | 26
  CS3: Yes | 4 | 2 | 4 | 10 | 9 | 8
  CS3: No | 13 | 13 | 8 | 7 | 7 | 18
  CS5: number analyzed (Participants) | 15 | 14 | 12 | 16 | 14 | 19
  CS5: Yes | 5 | 2 | 4 | 8 | 5 | 4
  CS5: No | 10 | 12 | 8 | 8 | 9 | 15
  CS6: number analyzed (Participants) | 17 | 14 | 10 | 16 | 17 | 23
  CS6: Yes | 6 | 3 | 1 | 10 | 4 | 6
  CS6: No | 11 | 11 | 9 | 6 | 13 | 17
  LTB: number analyzed (Participants) | 18 | 13 | 12 | 17 | 18 | 27
  LTB: Yes | 8 | 3 | 5 | 10 | 9 | 7
  LTB: No | 10 | 10 | 7 | 7 | 9 | 20

24. Secondary Outcome: Number and Percentage of 6-11 Month Old Subjects With ≥Four-fold Increase in Fecal Secretory Immunoglobulin A (SIgA) Response on Day 7, by Antigen
Description: as for outcome 23
Time Frame: 7 days
Population: Subjects who received both vaccinations and had valid baseline and endline immunologic samples.
Measure: Count of Participants; unit: Participants
Arm/Group | 6-11 Months: ETVAX (1/8) | 6-11 Months: ETVAX (1/4) | 6-11 Months: ETVAX (1/2) | 6-11 Months: ETVAX (1/4) + 2.5 ug dmLT | 6-11 Month Olds: ETVAX (1/4) + 5 ug dmLT | 6-11 Month Olds: Placebo
Number analyzed (Participants) | 23 | 23 | 16 | 20 | 21 | 37
Participants
  CFA/I: number analyzed (Participants) | 16 | 13 | 11 | 16 | 13 | 21
  CFA/I: Yes | 4 | 1 | 1 | 7 | 3 | 4
  CFA/I: No | 12 | 12 | 10 | 9 | 10 | 17
  CS3: number analyzed (Participants) | 17 | 15 | 12 | 17 | 16 | 26
  CS3: Yes | 2 | 0 | 1 | 6 | 2 | 2
  CS3: No | 15 | 15 | 11 | 11 | 14 | 24
  CS5: number analyzed (Participants) | 15 | 14 | 12 | 16 | 14 | 19
  CS5: Yes | 1 | 1 | 4 | 4 | 0 | 2
  CS5: No | 14 | 13 | 8 | 12 | 14 | 17
  CS6: number analyzed (Participants) | 17 | 14 | 10 | 16 | 17 | 23
  CS6: Yes | 3 | 0 | 1 | 7 | 1 | 5
  CS6: No | 14 | 14 | 9 | 9 | 16 | 18
  LTB: number analyzed (Participants) | 18 | 13 | 12 | 17 | 18 | 27
  LTB: Yes | 4 | 2 | 3 | 7 | 5 | 5
  LTB: No | 14 | 11 | 9 | 10 | 13 | 22

25. Secondary Outcome: Geometric Mean Titer (GMT) of Fecal Secretory Immunoglobulin A (SIgA) Response 6-11 Month Old Subjects on Day 7, by Antigen
Description: Fecal secretion was measured on Day 7 (7 days after administration of first dose of vaccine). Antigen in ETVAX were:
  E. coli, CFA/I, strain ETEX 21 formalin inactivated, E. coli, CS3, strain ETEX 22 formalin inactivated, E. coli, CS5, strain ETEX 23 formalin inactivated, E. coli, CS6, strain ETEX 24 phenol inactivated, B-subunit of the E. coli heat-labile enterotoxin
Time Frame: 7 days
Population: Subjects who received both vaccinations and had valid baseline and endline immunologic samples.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 6-11 Months: ETVAX (1/8) | 6-11 Months: ETVAX (1/4) | 6-11 Months: ETVAX (1/2) | 6-11 Months: ETVAX (1/4) + 2.5 ug dmLT | 6-11 Month Olds: ETVAX (1/4) + 5 ug dmLT | 6-11 Month Olds: Placebo
Number analyzed (Participants) | 23 | 23 | 16 | 20 | 21 | 37
titer
  CFA/I: number analyzed (Participants) | 16 | 13 | 11 | 16 | 13 | 21
  CFA/I | 49.6 [20.2 to 122] | 94.7 [35.7 to 251] | 53.8 [19.3 to 150] | 125 [59.8 to 260] | 70.6 [42.1 to 118] | 57.1 [28.7 to 114]
  CS3: number analyzed (Participants) | 17 | 15 | 12 | 17 | 16 | 26
  CS3 | 111 [45.4 to 270] | 94.7 [35.7 to 251] | 53.8 [19.3 to 150] | 125 [59.8 to 260] | 70.6 [42.1 to 118] | 57.1 [28.7 to 114]
  CS5: number analyzed (Participants) | 15 | 14 | 12 | 16 | 14 | 19
  CS5 | 27.8 [15.8 to 48.8] | 65 [30.9 to 137] | 19.5 [10.1 to 37.8] | 60.7 [37.1 to 99.3] | 59.8 [32.3 to 111] | 35.6 [22.3 to 56.9]
  CS6: number analyzed (Participants) | 17 | 14 | 10 | 10 | 17 | 23
  CS6 | 72 [39.7 to 130] | 80.7 [38.7 to 168] | 36.3 [20.1 to 65.6] | 187 [84.0 to 415] | 101 [62.7 to 164] | 101 [51.1 to 198]
  LTB: number analyzed (Participants) | 18 | 13 | 12 | 12 | 18 | 27
  LTB | 281 [154 to 511] | 474 [129 to 1747] | 345 [160 to 745] | 1249 [471 to 3311] | 536 [235 to 1219] | 448 [264 to 762]

26. Secondary Outcome: Geometric Mean Fold Change of Fecal Secretory Immunoglobulin A (SIgA) Response Among 6-11 Month Old Subjects on Day 7, by Antigen
Description: Fecal secretion was measured on Day 0 and Day 7 (7 days after administration of first dose of vaccine). Antigen in ETVAX were:
  E. coli, CFA/I, strain ETEX 21 formalin inactivated, E. coli, CS3, strain ETEX 22 formalin inactivated, E. coli, CS5, strain ETEX 23 formalin inactivated, E. coli, CS6, strain ETEX 24 phenol inactivated, B-subunit of the E. coli heat-labile enterotoxin
Time Frame: 7 days
Population: Subjects who received both vaccinations and had valid baseline and endline immunologic samples.
Measure: Geometric Mean (95% Confidence Interval); unit: fold change
Arm/Group | 6-11 Months: ETVAX (1/8) | 6-11 Months: ETVAX (1/4) | 6-11 Months: ETVAX (1/2) | 6-11 Months: ETVAX (1/4) + 2.5 ug dmLT | 6-11 Month Olds: ETVAX (1/4) + 5 ug dmLT | 6-11 Month Olds: Placebo
Number analyzed (Participants) | 23 | 23 | 16 | 20 | 21 | 37
fold change
  CFA/I: number analyzed (Participants) | 16 | 13 | 11 | 16 | 13 | 21
  CFA/I | 2.05 [1.16 to 3.63] | 0.98 [0.447 to 2.15] | 1.12 [0.418 to 3.02] | 2.92 [1.24 to 6.88] | 1.53 [0.708 to 3.29] | 1.07 [0.456 to 2.51]
  CS3: number analyzed (Participants) | 17 | 15 | 12 | 17 | 16 | 26
  CS3 | 1.32 [0.715 to 2.42] | 0.587 [0.373 to 0.925] | 0.884 [0.401 to 1.95] | 2.71 [1.11 to 6.64] | 1.73 [0.975 to 3.07] | 0.989 [0.613 to 1.60]
  CS5: number analyzed (Participants) | 15 | 14 | 12 | 16 | 14 | 19
  CS5 | 1.37 [0.900 to 2.09] | 0.981 [0.594 to 1.62] | 1.19 [0.496 to 2.85] | 2.22 [1.16 to 4.26] | 0.793 [0.383 to 1.64] | 0.841 [0.478 to 1.48]
  CS6: number analyzed (Participants) | 17 | 14 | 10 | 16 | 17 | 23
  CS6 | 1.09 [0.471 to 2.51] | 0.718 [0.424 to 1.22] | 0.529 [0.126 to 2.23] | 3.75 [1.51 to 9.32] | 1.02 [0.617 to 1.70] | 1.09 [0.479 to 2.49]
  LTB: number analyzed (Participants) | 18 | 13 | 12 | 17 | 18 | 27
  LTB | 1.63 [0.718 to 3.68] | 0.937 [0.523 to 1.68] | 1.76 [0.941 to 3.30] | 2.54 [1.06 to 6.09] | 2.01 [0.745 to 5.40] | 1.1 [0.601 to 2.03]

27. Secondary Outcome: Number and Percentage of 6-11 Month Old Subjects With ≥Two-fold Increase in Fecal Secretory Immunoglobulin A (SIgA) Response on Day 19, by Antigen
Description: Fecal secretion was measured on Day 0 and Day 19 (5 days after administration of second dose of vaccine). Antigen in ETVAX were:
  E. coli, CFA/I, strain ETEX 21 formalin inactivated, E. coli, CS3, strain ETEX 22 formalin inactivated, E. coli, CS5, strain ETEX 23 formalin inactivated, E. coli, CS6, strain ETEX 24 phenol inactivated, B-subunit of the E. coli heat-labile enterotoxin
Time Frame: Day 19
Population: Subjects who received both vaccinations and had valid baseline and endline immunologic samples.
Measure: Count of Participants; unit: Participants
Arm/Group | 6-11 Months: ETVAX (1/8) | 6-11 Months: ETVAX (1/4) | 6-11 Months: ETVAX (1/2) | 6-11 Months: ETVAX (1/4) + 2.5 ug dmLT | 6-11 Month Olds: ETVAX (1/4) + 5 ug dmLT | 6-11 Month Olds: Placebo
Number analyzed (Participants) | 23 | 23 | 16 | 20 | 21 | 37
Participants
  CFA/I: number analyzed (Participants) | 20 | 20 | 15 | 19 | 14 | 32
  CFA/I: Yes | 8 | 7 | 4 | 8 | 5 | 10
  CFA/I: No | 12 | 13 | 11 | 11 | 9 | 22
  CS3: number analyzed (Participants) | 21 | 22 | 16 | 20 | 18 | 35
  CS3: Yes | 5 | 7 | 5 | 7 | 8 | 9
  CS3: No | 16 | 15 | 11 | 13 | 10 | 26
  CS5: number analyzed (Participants) | 20 | 21 | 16 | 19 | 15 | 30
  CS5: Yes | 6 | 8 | 6 | 8 | 4 | 8
  CS5: No | 14 | 13 | 10 | 11 | 11 | 22
  CS6: number analyzed (Participants) | 20 | 22 | 14 | 19 | 18 | 33
  CS6: Yes | 6 | 7 | 4 | 8 | 5 | 8
  CS6: No | 14 | 15 | 10 | 11 | 13 | 25
  LTB: number analyzed (Participants) | 22 | 22 | 16 | 20 | 21 | 36
  LTB: Yes | 12 | 11 | 11 | 13 | 11 | 15
  LTB: No | 10 | 11 | 5 | 7 | 10 | 21

28. Secondary Outcome: Number and Percentage of 6-11 Month Old Subjects With ≥Four-fold Increase in Fecal Secretory Immunoglobulin A (SIgA) Response on Day 19, by Antigen
Description: Fecal secretion was measured on Day 0 and Day 19 (5 days after administration of second dose of vaccine). Antigens in ETVAX were:
  E. coli, CFA/I, strain ETEX 21 formalin inactivated, E. coli, CS3, strain ETEX 22 formalin inactivated, E. coli, CS5, strain ETEX 23 formalin inactivated, E. coli, CS6, strain ETEX 24 phenol inactivated, B-subunit of the E. coli heat-labile enterotoxin
Time Frame: 19 days
Population: Subjects who received both vaccinations and had valid baseline and endline immunologic samples.
Measure: Count of Participants; unit: Participants
Arm/Group | 6-11 Months: ETVAX (1/8) | 6-11 Months: ETVAX (1/4) | 6-11 Months: ETVAX (1/2) | 6-11 Months: ETVAX (1/4) + 2.5 ug dmLT | 6-11 Month Olds: ETVAX (1/4) + 5 ug dmLT | 6-11 Month Olds: Placebo
Number analyzed (Participants) | 23 | 23 | 16 | 20 | 21 | 37
Participants
  CFA/I: number analyzed (Participants) | 20 | 20 | 15 | 19 | 14 | 32
  CFA/I: Yes | 5 | 2 | 4 | 6 | 4 | 4
  CFA/I: No | 15 | 18 | 11 | 13 | 10 | 28
  CS3: number analyzed (Participants) | 21 | 22 | 16 | 20 | 18 | 35
  CS3: Yes | 2 | 4 | 3 | 5 | 3 | 3
  CS3: No | 19 | 18 | 13 | 15 | 15 | 32
  CS5: number analyzed (Participants) | 20 | 21 | 16 | 19 | 15 | 30
  CS5: Yes | 3 | 3 | 4 | 6 | 1 | 3
  CS5: No | 17 | 18 | 12 | 13 | 14 | 27
  CS6: number analyzed (Participants) | 20 | 22 | 14 | 19 | 18 | 33
  CS6: Yes | 0 | 5 | 2 | 6 | 1 | 7
  CS6: No | 20 | 17 | 12 | 13 | 17 | 26
  LTB: number analyzed (Participants) | 22 | 22 | 16 | 20 | 21 | 36
  LTB: Yes | 5 | 5 | 8 | 7 | 9 | 8
  LTB: No | 17 | 17 | 8 | 13 | 12 | 28

29. Secondary Outcome: Geometric Mean Titer (GMT) of Fecal Secretory Immunoglobulin A (SIgA) Response 6-11 Month Old Subjects on Day 19, by Antigen
Description: Fecal secretion was measured on Day 19 (5 days after administration of second dose of vaccine). Antigen in ETVAX were:
  E. coli, CFA/I, strain ETEX 21 formalin inactivated, E. coli, CS3, strain ETEX 22 formalin inactivated, E. coli, CS5, strain ETEX 23 formalin inactivated, E. coli, CS6, strain ETEX 24 phenol inactivated, B-subunit of the E. coli heat-labile enterotoxin
Time Frame: 19 days
Population: Subjects who received both vaccinations and had valid baseline and endline immunologic samples.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 6-11 Months: ETVAX (1/8) | 6-11 Months: ETVAX (1/4) | 6-11 Months: ETVAX (1/2) | 6-11 Months: ETVAX (1/4) + 2.5 ug dmLT | 6-11 Month Olds: ETVAX (1/4) + 5 ug dmLT | 6-11 Month Olds: Placebo
Number analyzed (Participants) | 23 | 23 | 16 | 20 | 21 | 37
titer
  CFA/I: number analyzed (Participants) | 20 | 20 | 15 | 19 | 21 | 32
  CFA/I | 37.3 [18.3 to 76.2] | 99.1 [57.6 to 170] | 40.2 [16.1 to 100] | 102 [50.2 to 209] | 48.9 [21.6 to 111] | 66.3 [43.7 to 100]
  CS3: number analyzed (Participants) | 21 | 22 | 16 | 20 | 21 | 35
  CS3 | 107 [47.8 to 240] | 158 [75.3 to 330] | 48.7 [17.1 to 139] | 136 [74.6 to 246] | 166 [94.9 to 292] | 118 [83.1 to 166]
  CS5: number analyzed (Participants) | 20 | 21 | 16 | 19 | 21 | 30
  CS5 | 27.8 [16.4 to 47.1] | 72.7 [40.1 to 132] | 22.1 [7.04 to 69.6] | 50.5 [34.3 to 74.3] | 63.5 [27.7 to 146] | 45.8 [33.0 to 63.4]
  CS6: number analyzed (Participants) | 20 | 22 | 14 | 19 | 21 | 33
  CS6 | 62.2 [33.2 to 117] | 135 [68.4 to 268] | 29.8 [11.5 to 77.7] | 121 [57.8 to 252] | 94.8 [60.0 to 150] | 110 [71.7 to 170]
  LTB: number analyzed (Participants) | 22 | 22 | 16 | 20 | 21 | 36
  LTB | 306 [171 to 549] | 1246 [627 to 2475] | 587 [202 to 1707] | 1507 [639 to 3559] | 838 [390 to 1802] | 533 [317 to 897]

30. Secondary Outcome: Geometric Mean Fold Change of Fecal Secretory Immunoglobulin A (SIgA) Response Among 6-11 Month Old Subjects on Day 19, by Antigen
Description: as for outcome 27
Time Frame: 19 days
Population: Subjects who received both vaccinations and had valid baseline and endline immunologic samples.
Measure: Geometric Mean (95% Confidence Interval); unit: fold change
Arm/Group | 6-11 Months: ETVAX (1/8) | 6-11 Months: ETVAX (1/4) | 6-11 Months: ETVAX (1/2) | 6-11 Months: ETVAX (1/4) + 2.5 ug dmLT | 6-11 Month Olds: ETVAX (1/4) + 5 ug dmLT | 6-11 Month Olds: Placebo
Number analyzed (Participants) | 23 | 23 | 16 | 20 | 21 | 37
fold change
  CFA/I: number analyzed (Participants) | 20 | 20 | 15 | 19 | 14 | 32
  CFA/I | 1.81 [1.12 to 2.91] | 1.18 [0.627 to 2.23] | 0.975 [0.292 to 3.25] | 2.31 [1.16 to 4.59] | 1.08 [0.366 to 3.18] | 1.23 [0.780 to 1.94]
  CS3: number analyzed (Participants) | 21 | 22 | 16 | 20 | 18 | 35
  CS3 | 1.36 [0.946 to 1.94] | 1.19 [0.641 to 2.22] | 0.97 [0.310 to 3.04] | 1.88 [0.923 to 3.84] | 1.52 [0.820 to 2.80] | 1.1 [0.754 to 1.61]
  CS5: number analyzed (Participants) | 20 | 21 | 16 | 19 | 15 | 30
  CS5 | 1.44 [0.848 to 2.44] | 1.24 [0.599 to 2.58] | 1.37 [0.423 to 4.44] | 1.92 [0.991 to 3.71] | 0.888 [0.408 to 1.93] | 1.1 [0.710 to 1.72]
  CS6: number analyzed (Participants) | 20 | 22 | 14 | 19 | 18 | 33
  CS6 | 0.896 [0.529 to 1.52] | 1.42 [0.655 to 3.07] | 0.457 [0.109 to 1.92] | 2.41 [1.09 to 5.32] | 0.96 [0.533 to 1.73] | 1.2 [0.739 to 1.94]
  LTB: number analyzed (Participants) | 22 | 22 | 16 | 20 | 21 | 36
  LTB | 1.75 [0.809 to 3.77] | 1.99 [0.987 to 4.00] | 3.25 [1.03 to 10.2] | 3.19 [1.52 to 6.69] | 3.64 [1.45 to 9.12] | 1.64 [0.904 to 2.96]

31. Secondary Outcome: Number and Percentage of 6-11 Month Old Subjects With ≥Two-fold Increase in Fecal Secretory Immunoglobulin A (SIgA) Response on Day 28, by Antigen
Description: Fecal secretion was measured on Day 0 and Day 28 (2 weeks after administration of second dose of vaccine). Antigen in ETVAX were:
  E. coli, CFA/I, strain ETEX 21 formalin inactivated, E. coli, CS3, strain ETEX 22 formalin inactivated, E. coli, CS5, strain ETEX 23 formalin inactivated, E. coli, CS6, strain ETEX 24 phenol inactivated, B-subunit of the E. coli heat-labile enterotoxin
Time Frame: 28 days
Population: Subjects who received both vaccinations and had valid baseline and endline immunologic samples.
Measure: Count of Participants; unit: Participants
Arm/Group | 6-11 Months: ETVAX (1/8) | 6-11 Months: ETVAX (1/4) | 6-11 Months: ETVAX (1/2) | 6-11 Months: ETVAX (1/4) + 2.5 ug dmLT | 6-11 Month Olds: ETVAX (1/4) + 5 ug dmLT | 6-11 Month Olds: Placebo
Number analyzed (Participants) | 23 | 23 | 16 | 20 | 21 | 37
Participants
  CFA/I: number analyzed (Participants) | 12 | 16 | 11 | 18 | 9 | 26
  CFA/I: Yes | 7 | 6 | 5 | 10 | 5 | 10
  CFA/I: No | 5 | 10 | 6 | 8 | 4 | 16
  CS3: number analyzed (Participants) | 15 | 16 | 12 | 19 | 12 | 27
  CS3: Yes | 5 | 4 | 5 | 11 | 8 | 14
  CS3: No | 10 | 12 | 7 | 8 | 4 | 13
  CS5: number analyzed (Participants) | 13 | 16 | 12 | 18 | 8 | 23
  CS5: Yes | 5 | 4 | 4 | 9 | 3 | 5
  CS5: No | 8 | 12 | 8 | 9 | 5 | 18
  CS6: number analyzed (Participants) | 14 | 16 | 10 | 18 | 9 | 25
  CS6: Yes | 5 | 7 | 3 | 10 | 4 | 6
  CS6: No | 9 | 9 | 7 | 8 | 5 | 19
  LTB: number analyzed (Participants) | 16 | 15 | 12 | 19 | 14 | 28
  LTB: Yes | 8 | 8 | 10 | 12 | 9 | 10
  LTB: No | 8 | 7 | 2 | 7 | 5 | 18

32. Secondary Outcome: Number and Percentage of 6-11 Month Old Subjects With ≥Four-fold Increase in Fecal Secretory Immunoglobulin A (SIgA) Response on Day 28, by Antigen
Description: Fecal secretion was measured on Day 0 and Day 28 (2 weeks after administration of second dose of vaccine). Antigens in ETVAX were:
  E. coli, CFA/I, strain ETEX 21 formalin inactivated, E. coli, CS3, strain ETEX 22 formalin inactivated, E. coli, CS5, strain ETEX 23 formalin inactivated, E. coli, CS6, strain ETEX 24 phenol inactivated, B-subunit of the E. coli heat-labile enterotoxin
Time Frame: 28 days
Population: Subjects who received both vaccinations and had valid baseline and endline immunologic samples.
Measure: Count of Participants; unit: Participants
Arm/Group | 6-11 Months: ETVAX (1/8) | 6-11 Months: ETVAX (1/4) | 6-11 Months: ETVAX (1/2) | 6-11 Months: ETVAX (1/4) + 2.5 ug dmLT | 6-11 Month Olds: ETVAX (1/4) + 5 ug dmLT | 6-11 Month Olds: Placebo
Number analyzed (Participants) | 23 | 23 | 16 | 20 | 21 | 37
Participants
  CFA/I: number analyzed (Participants) | 12 | 16 | 11 | 18 | 9 | 26
  CFA/I: Yes | 4 | 4 | 4 | 6 | 5 | 4
  CFA/I: No | 8 | 12 | 7 | 12 | 4 | 22
  CS3: number analyzed (Participants) | 15 | 16 | 12 | 19 | 12 | 27
  CS3: Yes | 2 | 4 | 1 | 6 | 5 | 8
  CS3: No | 13 | 12 | 11 | 13 | 7 | 19
  CS5: number analyzed (Participants) | 13 | 16 | 12 | 18 | 8 | 23
  CS5: Yes | 3 | 3 | 4 | 7 | 1 | 3
  CS5: No | 10 | 13 | 8 | 11 | 7 | 20
  CS6: number analyzed (Participants) | 14 | 16 | 10 | 18 | 9 | 25
  CS6: Yes | 3 | 4 | 2 | 7 | 2 | 4
  CS6: No | 11 | 12 | 8 | 11 | 7 | 21
  LTB: number analyzed (Participants) | 16 | 15 | 12 | 19 | 14 | 28
  LTB: Yes | 7 | 5 | 6 | 11 | 7 | 7
  LTB: No | 9 | 10 | 6 | 8 | 7 | 21

33. Secondary Outcome: Geometric Mean Titer (GMT) of Fecal Secretory Immunoglobulin A (SIgA) Response 6-11 Month Old Subjects on Day 28, by Antigen
Description: Fecal secretion was measured on Day 28 (2 weeks after administration of second dose of vaccine). Antigen in ETVAX were:
  E. coli, CFA/I, strain ETEX 21 formalin inactivated, E. coli, CS3, strain ETEX 22 formalin inactivated, E. coli, CS5, strain ETEX 23 formalin inactivated, E. coli, CS6, strain ETEX 24 phenol inactivated, B-subunit of the E. coli heat-labile enterotoxin
Time Frame: 28 days
Population: Subjects who received both vaccinations and had valid baseline and endline immunologic samples.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 6-11 Months: ETVAX (1/8) | 6-11 Months: ETVAX (1/4) | 6-11 Months: ETVAX (1/2) | 6-11 Months: ETVAX (1/4) + 2.5 ug dmLT | 6-11 Month Olds: ETVAX (1/4) + 5 ug dmLT | 6-11 Month Olds: Placebo
Number analyzed (Participants) | 23 | 23 | 16 | 20 | 21 | 37
titer
  CFA/I: number analyzed (Participants) | 12 | 16 | 11 | 18 | 9 | 26
  CFA/I | 52.4 [18.4 to 149] | 178 [76.7 to 414] | 72.6 [22.2 to 237] | 126 [57.6 to 274] | 136 [90.9 to 204] | 61.8 [34.4 to 111]
  CS3: number analyzed (Participants) | 15 | 16 | 12 | 19 | 12 | 27
  CS3 | 106 [40.1 to 281] | 271 [105 to 699] | 57.5 [32.6 to 101] | 223 [120 to 413] | 373 [158 to 877] | 181 [121 to 273]
  CS5: number analyzed (Participants) | 13 | 16 | 12 | 18 | 8 | 23
  CS5 | 28.8 [15.4 to 281] | 271 [105 to 699] | 57.5 [32.6 to 101] | 223 [120 to 413] | 373 [158 to 877] | 181 [121 to 273]
  CS6: number analyzed (Participants) | 14 | 16 | 10 | 18 | 9 | 25
  CS6 | 57.8 [29.0 to 115] | 145 [72.2 to 293] | 44.2 [13.0 to 150] | 138 [71.8 to 266] | 163 [55.3 to 484] | 86.1 [45.8 to 162]
  LTB: number analyzed (Participants) | 16 | 15 | 12 | 19 | 14 | 28
  LTB | 517 [264 to 1010] | 2151 [875 to 5291] | 911 [364 to 2277] | 2231 [1018 to 4888] | 1128 [376 to 3381] | 391 [230 to 665]

34. Secondary Outcome: Geometric Mean Fold Change of Fecal Secretory Immunoglobulin A (SIgA) Response Among 6-11 Month Old Subjects on Day 28, by Antigen
Description: as for outcome 31
Time Frame: 28 days
Population: Subjects who received both vaccinations and had valid baseline and endline immunologic samples.
Measure: Geometric Mean (95% Confidence Interval); unit: fold change
Arm/Group | 6-11 Months: ETVAX (1/8) | 6-11 Months: ETVAX (1/4) | 6-11 Months: ETVAX (1/2) | 6-11 Months: ETVAX (1/4) + 2.5 ug dmLT | 6-11 Month Olds: ETVAX (1/4) + 5 ug dmLT | 6-11 Month Olds: Placebo
Number analyzed (Participants) | 23 | 23 | 16 | 20 | 21 | 37
fold change
  CFA/I: number analyzed (Participants) | 12 | 16 | 11 | 18 | 9 | 26
  CFA/I | 2.74 [1.16 to 6.47] | 2.35 [0.930 to 5.92] | 1.46 [0.380 to 5.92] | 2.73 [1.18 to 6.34] | 2.35 [0.941 to 5.88] | 1.32 [0.767 to 2.28]
  CS3: number analyzed (Participants) | 15 | 16 | 12 | 19 | 12 | 27
  CS3 | 1.28 [0.512 to 3.20] | 1.59 [0.528 to 4.81] | 1.02 [0.408 to 2.55] | 2.83 [1.33 to 6.04] | 3.08 [1.69 to 5.61] | 1.71 [1.02 to 2.86]
  CS5: number analyzed (Participants) | 13 | 16 | 12 | 18 | 8 | 23
  CS5 | 1.63 [0.857 to 3.10] | 1.61 [0.757 to 3.42] | 1.42 [0.410 to 4.91] | 1.85 [0.929 to 3.70] | 1.18 [0.484 to 2.87] | 1.16 [0.618 to 2.17]
  CS6: number analyzed (Participants) | 14 | 16 | 10 | 18 | 9 | 25
  CS6 | 0.882 [0.401 to 1.94] | 1.5 [0.723 to 3.10] | 0.709 [0.180 to 2.80] | 2.6 [1.32 to 5.15] | 1.39 [0.593 to 3.24] | 1.05 [0.575 to 1.93]
  LTB: number analyzed (Participants) | 16 | 15 | 16 | 19 | 19 | 28
  LTB | 2.14 [0.763 to 6.01] | 1.92 [0.755 to 4.90] | 4.58 [1.79 to 11.7] | 5.33 [2.01 to 14.2] | 4.65 [1.41 to 15.3] | 1.19 [0.612 to 2.31]

ADVERSE EVENTS:
Time Frame: 6 months ± 14 days after the first dose for unsolicited adverse events, 7 days for solicited events (fever, vomiting, loose stools, diarrhea, acute systemic allergic reaction; plus nausea and abdominal pain/stomach ache for adults/children 24-59 months)
Arm/Group | Adult: ETVAX (Full) | Adult: ETVAX (Full) + 10 ug dmLT | Adult: Placebo | 24-59 Months: ETVAX (1/4) | 24-59 Months: ETVAX (1/2) | 24-59 Months: ETVAX (Full) | 24-59 Months: ETVAX (1/2) + 2.5 ug dmLT | 24-59 Months: ETVAX (1/2) + 5 ug dmLT | 24-59 Months: ETVAX (1/2) + 10 ug dmLT | 24-59 Months: Placebo | 12-23 Months: ETVAX (1/4) | 12-23 Months: ETVAX (1/2) | 12-23 Months: ETVAX (1/2) + 2.5 ug dmLT | 12-23 Months: ETVAX (1/2) + 5 ug dmLT | 12-23 Months: Placebo | 6-11 Months: ETVAX (1/8) | 6-11 Months: ETVAX (1/4) | 6-11 Months: ETVAX (1/2) | 6-11 Months: ETVAX (1/4) + 2.5 ug dmLT | 6-11 Month Olds: ETVAX (1/4) + 5 ug dmLT | 6-11 Month Olds: Placebo
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15 | 0/15 | 0/3 | 0/15 | 0/15 | 0/15 | 0/52 | 0/15 | 0/15 | 0/15 | 0/15 | 0/40 | 0/30 | 0/30 | 0/30 | 0/30 | 0/30 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15 | 0/15 | 0/3 | 0/15 | 0/15 | 0/15 | 1/52 | 1/15 | 0/15 | 0/15 | 0/15 | 0/40 | 0/30 | 0/30 | 1/30 | 0/30 | 0/30 | 0/50
Other Adverse Events (participants affected / at risk) | 0/15 | 4/15 | 1/15 | 2/15 | 1/15 | 2/3 | 4/15 | 1/15 | 3/15 | 4/52 | 5/15 | 2/15 | 6/15 | 9/15 | 5/40 | 4/30 | 8/30 | 13/30 | 9/30 | 8/30 | 10/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adult: ETVAX (Full) (N=15) | Adult: ETVAX (Full) + 10 ug dmLT (N=15) | Adult: Placebo (N=15) | 24-59 Months: ETVAX (1/4) (N=15) | 24-59 Months: ETVAX (1/2) (N=15) | 24-59 Months: ETVAX (Full) (N=3) | 24-59 Months: ETVAX (1/2) + 2.5 ug dmLT (N=15) | 24-59 Months: ETVAX (1/2) + 5 ug dmLT (N=15) | 24-59 Months: ETVAX (1/2) + 10 ug dmLT (N=15) | 24-59 Months: Placebo (N=52) | 12-23 Months: ETVAX (1/4) (N=15) | 12-23 Months: ETVAX (1/2) (N=15) | 12-23 Months: ETVAX (1/2) + 2.5 ug dmLT (N=15) | 12-23 Months: ETVAX (1/2) + 5 ug dmLT (N=15) | 12-23 Months: Placebo (N=40) | 6-11 Months: ETVAX (1/8) (N=30) | 6-11 Months: ETVAX (1/4) (N=30) | 6-11 Months: ETVAX (1/2) (N=30) | 6-11 Months: ETVAX (1/4) + 2.5 ug dmLT (N=30) | 6-11 Month Olds: ETVAX (1/4) + 5 ug dmLT (N=30) | 6-11 Month Olds: Placebo (N=50)
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rickets (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adult: ETVAX (Full) (N=15) | Adult: ETVAX (Full) + 10 ug dmLT (N=15) | Adult: Placebo (N=15) | 24-59 Months: ETVAX (1/4) (N=15) | 24-59 Months: ETVAX (1/2) (N=15) | 24-59 Months: ETVAX (Full) (N=3) | 24-59 Months: ETVAX (1/2) + 2.5 ug dmLT (N=15) | 24-59 Months: ETVAX (1/2) + 5 ug dmLT (N=15) | 24-59 Months: ETVAX (1/2) + 10 ug dmLT (N=15) | 24-59 Months: Placebo (N=52) | 12-23 Months: ETVAX (1/4) (N=15) | 12-23 Months: ETVAX (1/2) (N=15) | 12-23 Months: ETVAX (1/2) + 2.5 ug dmLT (N=15) | 12-23 Months: ETVAX (1/2) + 5 ug dmLT (N=15) | 12-23 Months: Placebo (N=40) | 6-11 Months: ETVAX (1/8) (N=30) | 6-11 Months: ETVAX (1/4) (N=30) | 6-11 Months: ETVAX (1/2) (N=30) | 6-11 Months: ETVAX (1/4) + 2.5 ug dmLT (N=30) | 6-11 Month Olds: ETVAX (1/4) + 5 ug dmLT (N=30) | 6-11 Month Olds: Placebo (N=50)
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bronchiolitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dandruff (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Foreign body in eye (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Keratitis (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Measles (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Varicella (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 2 | 1 | 0 | 3 | 1 | 1 | 2 | 2 | 2 | 3 | 3 | 6
Vomiting (General disorders) | 0 | 0 | 0 | 2 | 0 | 2 | 2 | 1 | 3 | 0 | 2 | 1 | 2 | 8 | 0 | 2 | 5 | 8 | 6 | 5 | 2
Loose stools (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 3 | 1 | 0 | 1 | 3 | 2 | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-06-01): https://cdn.clinicaltrials.gov/large-docs/02/NCT02531802/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-08): https://cdn.clinicaltrials.gov/large-docs/02/NCT02531802/SAP_001.pdf